# CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN for DMID Protocol: 14-0015 Study Title:

A Phase II Study to Evaluate and Compare the Immunogenicity of Monovalent Inactivated Influenza A/H7N9 Virus Vaccine Administered with and without AS03 Adjuvant and Monovalent Inactivated Influenza A/H3N2v Virus Vaccine Administered without Adjuvant in Healthy Adults through Standard and Systems Biology Analyses

NCT02921997

Version 1.0

**DATE: 21 NOVEMBER 2019** 

THIS COMMUNICATION IS PRIVILEGED AND CONFIDENTIAL

# **STUDY TITLE**

| <b>Protocol Number Code:</b> | DMID Protocol: 14-0015 |
|---|---|
| <b>Development Phase:</b> | Phase II |
| Products: | Monovalent Inactivated Influenza A/Shanghai/02/2013 (H7N9) Virus Vaccine Administered with and without AS03 Adjuvant |
| | Monovalent Inactivated Influenza A/Minnesota/11/2010 (H3N2)v Virus Vaccine Administered without Adjuvant |
| Form/Route: | Intramuscular |
| Indication Studied: | Influenza |
| Sponsor: | Division of Microbiology and Infectious Diseases |
| | National Institute of Allergy and Infectious Diseases |
| | National Institutes of Health |
| Clinical Trial Initiation Date: | 01 November 2016 |
| Clinical Trial Completion Date: | 14 February 2018 |
| Date of the Analysis Plan: | 21 November 2019 |
| Version Number: | 1.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# TABLE OF CONTENTS

| STUDY | TITLE | II |
|---|---|---|
| TABLE | OF CONTENTS | III |
| LIST OF | F ABBREVIATIONS | VI |
| 1. | PREFACE | 1 |
| 2. | INTRODUCTION | 2 |
| 2.1. | Purpose of the Analyses | 2 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 3 |
| 3.1. | Study Objectives | 3 |
| 3.2. | Endpoints | 4 |
| 3.3. | Study Definitions and Derived Variables | 6 |
| 4. | INVESTIGATIONAL PLAN | 7 |
| 4.1. | Overall Study Design and Plan | 7 |
| 4.2. | Discussion of Study Design, Including the Choice of Control Groups | 8 |
| 4.3. | Selection of Study Population | 8 |
| 4.4. | Treatments | 11 |
| 4.4.1. | Treatments Administered. | 11 |
| 4.4.2. | Identity of Investigational Product(s) | 12 |
| 4.4.3. | Method of Assigning Subjects to Treatment Groups (Randomization) | 12 |
| 4.4.4. | Selection of Doses in the Study | 13 |
| 4.4.5. | Selection and Timing of Dose for Each Subject | 13 |
| 4.4.6. | Blinding | 13 |
| 4.4.7. | Prior and Concomitant Therapy | 13 |
| 4.4.8. | Treatment Compliance | 14 |
| 4.5. | Immunogenicity and Safety Variables | 14 |
| 4.5.1. | Immunogenicity Variables | 14 |
| 4.5.2. | -Omics Variables | 14 |
| 4.5.3. | Safety Variables | 15 |
| 5. | SAMPLE SIZE CONSIDERATIONS | 16 |
| 6. | GENERAL STATISTICAL CONSIDERATIONS | 17 |
| 6.1. | General Principles | 17 |

# **Table of Contents** (continued)

| 6.2. | Timing of Analyses | 17 |
|---|---|---|
| 6.3. | Analysis Populations | |
| 6.3.1. | Safety Analysis Population | 17 |
| 6.3.2. | Intention-to-Treat Analysis (ITT) Population | 17 |
| 6.3.3. | Per protocol (PP) Population | 17 |
| 6.3.4. | The -Omics Analysis Population | |
| 6.4. | Covariates and Subgroups | |
| 6.5. | Missing Data | |
| 6.6. | Interim Analyses and Data Monitoring | 18 |
| 6.7. | Multicenter Studies | 18 |
| 6.8. | Multiple Comparisons/Multiplicity | 18 |
| 7. | STUDY SUBJECTS | 19 |
| 7.1. | Disposition of Subjects | 19 |
| 7.2. | Protocol Deviations | 19 |
| 8. | IMMUNOGENICITY EVALUATION | 20 |
| 8.1. | Serum Antibody Analysis | 20 |
| 8.2. | Plasma Cytokines/Chemokine Analysis | 20 |
| 9. | TRANSCRIPTOMICS EVALUATIONS | 21 |
| 9.1. | RNA-Seq Data Processing and Qc | 21 |
| 9.1.1. | Human Reference Genome Alignment and Quality Assessment | 21 |
| 9.1.2. | Gene Expression Quantification and Data Normalization | 21 |
| 9.1.3. | Global Outlier and Batch Effect Detection | 21 |
| 9.1.4. | Pre-Vaccination Transcriptomics Activity | 22 |
| 9.1.5. | Log Fold Change Calculations | 22 |
| 9.1.6. | Determination of Cut Offs for Filtering Lowly Expressed Genes | 22 |
| 9.2. | Identification of Differentially Expressed Genes | 22 |
| 9.2.1. | Identification of DE Genes Compared to Pre-First Vaccination | 23 |
| 9.2.2. | Identification of DE Genes Compared to Pre-Second Vaccination | 23 |
| 9.2.3. | Identification of Genes with Differential Responses Between Study Arms | |
| 9.3. | Determination of higher order functional and temporal organization of differentially expressed genes | 24 |
| 9.3.1. | Subject-level Response Heatmaps | 24 |

# **Table of Contents** (continued)

| 9.3.2. | Identification of Co-Expressed Gene Clusters | 24 |
|---|---|---|
| 9.3.3. | Pathway Enrichment Analysis | 24 |
| 9.3.4. | Protein-Protein Interactions Network Analysis | 25 |
| 10. | SAFETY EVALUATIONS | 26 |
| 10.1. | Demographic and Other Baseline Characteristics | |
| 10.2. | Adverse Events | 26 |
| 10.2.1. | Solicited Events and Symptoms | 26 |
| 10.2.2. | Unsolicited Adverse Events | 26 |
| 10.3. | Deaths, Serious Adverse Events and other Significant Adverse Events | 27 |
| 10.4. | Vital Signs and Physical Evaluations | 27 |
| 11. | TERTIARY AND EXPLORATORY PROTEOMICS ANALYSES | 28 |
| 12. | EXPLORATORY CORRELATION ANALYSES | 29 |
| 13. | REPORTING CONVENTIONS | 30 |
| 14. | REFERENCES | 31 |
| 15. | LISTING OF TABLES, FIGURES, AND LISTINGS | 32 |
| APPEND | DICES | 33 |
| APPEND | IX 1. TABLE MOCK-UPS | 34 |
| APPEND | IX 2. FIGURE MOCK-UPS | 92 |
| APPEND | DIX 3 LISTINGS MOCK-UPS | 107 |

# LIST OF ABBREVIATIONS

| A/H3N2v | Influenza A Virus of the H3N2 Variant Subtype |
|---|---|
| A/H5N1 | Influenza A Virus of the H5N1 Subtype |
| A/H7N9 | Influenza A Virus of the H7N9 Subtype |
| AdvantageEDCSM | Electronic Data Capture System |
| AE | Adverse Event/Adverse Experience |
| AS03 | Adjuvant System (03) |
| α | Alpha |
| BMI | Body Mass Index |
| BPM | Beats Per Minute |
| CDC | Centers for Disease Control and Prevention |
| CDF | Cumulative Distribution Function |
| CI | Confidence Interval |
| CSR | Clinical Study Report |
| °C | Degrees Celsius |
| °F | Degrees Fahrenheit |
| D | Day(s) |
| DE | Differentially Expressed |
| DHHS | Department of Health and Human Services |
| DMID | Division of Microbiology and Infectious Diseases, NIAID, NIH |
| eCRF | Electronic Case Report Form |
| ESR | Erythrocyte Sedimentation Rate |
| FDA | Food and Drug Administration |
| FDR | False-discovery Rate |
| GCP | Good Clinical Practice |
| GMT | Geometric Mean Titer |
| GTF | Gene Transfer Format |
| HA | Hemagglutinin |
| HAI | Hemagglutination Inhibition |
| HIV | Human Immunodeficiency Virus |
| ICH | International Conference on Harmonisation |
| IFN | Interferon |
| IL | Interleukin |
| IM | Intramuscular |
| IQR | Interquartile Range |
| ITT | Intent-to-Treat |
| LCPM | Log2 Counts per Million |
| LFC | Log <sub>2</sub> Fold Change |
| LOD | Limit of Detection |
| MAAEs | Medically-Attended Adverse Events |
| mcg or µg | Microgram(s) |
| MedDRA® | Medical Dictionary for Regulatory Activities |

| mL | Milliliter(s) |
|---|---|
| mm | Millimeter(s) |
| mmHg | Millimeters of Mercury |
| MOP | Manual of Procedures |
| N | Number of Subjects |
| Neut or NT | Neutralizing or Neutralization |
| NIAID | National Institute of Allergy and Infectious Diseases, NIH, DHHS |
| NK | Natural Killer |
| NIH | National Institutes of Health |
| NOCMCs | New-Onset Chronic Medical Conditions |
| PBS | Phosphate-Buffered Saline |
| PIMMCs | Potentially Immune-Mediated Medical Conditions |
| PP | Per Protocol |
| QC | Quality Control |
| RCDF | Reverse Cumulative Distribution Function |
| RNA | Ribonucleic Acid |
| RP-HPLC | Reversed-Phase High-Performance Liquid Chromatography |
| SAE | Serious Adverse Event/Serious Adverse Experience |
| SAP | Statistical Analysis Plan |
| SDCC | Statistical and Data Coordinating Center |
| SOC | System Organ Class |
| SRID | Single Radial Immunodiffusion |
| TMM | Trimmed Mean of M-values |
| TNF | Tumor Necrosis Factor |
| US | United States |
| V | Visit(s) |
| VTEU | Vaccine and Treatment Evaluation Unit |
| WHO | World Health Organization |

#### 1. PREFACE

The Statistical Analysis Plan (SAP) for "A Phase II Study to Evaluate and Compare the Immunogenicity of Monovalent Inactivated Influenza A/H7N9 Virus Vaccine Administered with and without AS03 Adjuvant and Monovalent Inactivated Influenza A/H3N2v Virus Vaccine Administered without Adjuvant in Healthy Adults through Standard and Systems Biology Analyses" (DMID Protocol 14-0015) describes and expands upon the statistical information presented in the protocol.

This document describes all planned analyses including sample tables, listings, and figures. Regarding the final analyses and Clinical Study Report (CSR), this SAP follows the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice.

This document contains four sections: (1) a review of the study design, (2) general statistical considerations, (3) comprehensive statistical analysis methods for immunogenicity, transcriptomics, cytokine/chemokine, and safety outcomes, and (4) a list of proposed tables, figures, and listings. Within the table, figure, and listing mock-ups (Appendices 1, 2, and 3), references to CSR sections are included. Any deviation from this SAP will be described and justified in protocol amendments and/or in the CSR, as appropriate. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments. Tertiary and exploratory proteomics assessments and correlation analyses are presented in a separate addendum to this SAP.

# 2. INTRODUCTION

# 2.1. Purpose of the Analyses

The primary goal of these analyses is to characterize and compare gene expression responses from subjects receiving two doses of monovalent inactivated influenza A/Shanghai/02/2013 (H7N9) virus vaccine, hereafter referred to as A/H7N9 vaccine, administered with AS03 adjuvant with those subjects that received the same vaccine without AS03 post first and second dose. This direct comparison will potentially reveal gene expression signatures that are modulated by AS03 which in turn could lead to a better understanding of the immune response-enhancing capabilities of the AS03 adjuvant. As a co-primary endpoint, anti-HA hemagglutination-inhibition (HAI) antibody responses will be assessed. The secondary endpoint analysis focuses on serum neutralizing antibodies and plasma cytokine/chemokine profiles pre- and post-vaccination. As part of the tertiary analysis, A/H7N9 transcriptomics responses will be compared to a control arm receiving one dose of monovalent inactivated influenza A/Minnesota/11/2010 (H3N2)v virus vaccine, hereafter referred to as A/H3N2v vaccine. The goal is to compare the innate and adaptive immune responses observed between the two avian (A/H7N9) study arms, and between the unadjuvanted avian (A/H7N9) and a swine-origin influenza vaccine (A/H3N2v) that is more similar to seasonal influenza A/H3N2.

Additional tertiary and exploratory endpoint analyses are aimed at characterizing and comparing proteomics signatures and assessing the correlation between omics and serum antibody and plasma cytokines/chemokines as well as safety outcomes. The goal of the correlation analysis is to integrate the different data to develop a systems model of the human immune response to unadjuvanted monovalent inactivated influenza A/H3N2v virus vaccine and monovalent inactivated influenza A/H7N9 virus vaccine given with and without AS03 adjuvant.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

# 3.1. Study Objectives

# **Primary Objectives**

- 1. To assess the serum anti-HA hemagglutination-inhibition (HAI) response to influenza A/H7N9 antigen (with and without adjuvant) at Day 57 (approximately one month after the second study vaccination with A/H7N9 vaccine ± AS03) and influenza A/H3N2v antigen at Day 29 (approximately one month after the study vaccination with A/H3N2v vaccine).
- 2. To identify differentially expressed genes in human immune cells on Days 2, 4, and 29 (following the first study vaccination with A/H7N9 vaccine ± AS03) and on Days 30, 32, and 36 (following the second study vaccination with A/H7N9 vaccine ± AS03), compared to baseline assessments performed prior to each study vaccination (Days -7, 1, and 29).

# **Secondary Objectives**

- 1. To compare plasma cytokine and chemokine profiles at specific time points and between treatment arms:
  - a. Post-vaccination time points [(Days 2 and 4; Day 8 (A/H3N2v arm only)], and Days 30, 32, and 36 (A/H7N9 arms only) with pre-vaccination time points (Days -7 and 1, prior to first study vaccination and Day 29, prior to second study vaccination (A/H7N9 arms only).
- 2. To assess the neutralizing antibody responses to influenza A/H7N9 antigen (with and without adjuvant) at Day 57 (approximately one month after the second study vaccination with A/H7N9 vaccine ± AS03) and influenza A/H3N2v antigen at Day 29 (approximately one month after the study vaccination with A/H3N2v vaccine).
- 3. To identify differentially expressed genes in human immune cells on Days 2, 4, and 8 following one intramuscular dose of influenza A/H3N2v vaccine compared to baseline assessments performed prior to study vaccination (Day -7 and Day 1).

# **Tertiary Objectives**

- 1. To assess the frequency of adverse events.
- 2. To identify differentially abundant cellular proteins in human immune cells on Days 2, 4, and 8 following one intramuscular dose of influenza A/H3N2v vaccine compared to baseline assessments performed prior to study vaccination (Day -7 and Day 1).
- 3. To identify differentially abundant cellular proteins in human immune cells on Days 2, 4, and 29 (following first study vaccination with A/H7N9 vaccine ± AS03) and Days 30, 32, and 36 (following second study vaccination with A/H7N9 vaccine ± AS03), compared to baseline assessments performed prior to study vaccination (Days -7, 1, and 29).

# **Exploratory Objectives**

1. To identify and characterize differentially expressed genes in human immune cells on Days 2, 4, and 29 (following the first study vaccination with A/H7N9 vaccine ± AS03) and on Days 30, 32, and 36 (following the second study vaccination with A/H7N9 vaccine ± AS03) that differ between treatments (A/H7N9 vaccine vs. A/H7N9 vaccine + AS03).

- 2. To identify and characterize differentially abundant cellular proteins in human immune cells on Days 2, 4, and 29 (following the first study vaccination with A/H7N9 vaccine ± AS03) and on Days 30, 32, and 36 (following the second study vaccination with A/H7N9 vaccine ± AS03) that differ between treatments (A/H7N9 vaccine vs. A/H7N9 vaccine + AS03).
- 3. To identify and characterize differentially expressed genes in human immune cells on Days 2 and 4 (following the first study vaccination) that differ in baseline responses (Days -7, and 1) between treatments (A/H3N2v vaccine vs. A/H7N9 vaccine and A/H3N2v vaccine vs. A/H7N9 vaccine + AS03).
- 4. To identify and characterize differentially abundant cellular proteins in human immune cells on Days 2 and 4 (following the first study vaccination) that differ in baseline responses (Days -7, and 1) between treatments (A/H3N2v vaccine vs. A/H7N9 vaccine and A/H3N2v vaccine vs. A/H7N9 vaccine + AS03).
- 5. To identify transcriptomic and proteomic signatures in human immune cells that correlate with influenza seroconversion and with peak HAI titers.
- 6. To correlate plasma cytokine profiles with transcriptomic and proteomic profiles in subjects receiving influenza A/H3N2v vaccine or influenza A/H7N9 ± AS03 vaccine.
- 7. Exploratory inspection of transcriptomics\proteomics response signatures for subjects with unexpected or severe safety profiles that are related to the study products.

# 3.2. Endpoints

# **Primary Endpoints**

- 1. Percentage of subjects achieving seroconversion (defined as either a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer ≥1:40 or a pre- vaccination HAI titer ≥1:10 and a minimum four-fold rise in post-vaccination HAI antibody titer) at approximately 28 days after the second study vaccination (A/H7N9 vaccine, with and without adjuvant).
- 2. Percentage of subjects achieving seroconversion at approximately 28 days after the study vaccination with A/H3N2v vaccine.
- 3. Number of differentially expressed genes based on RNA expression as determined by RNA-Seq analysis, in human immune cells at Days 2, 4, 29, 30, 32, and 36 after study vaccination with AS03-adjuvanted and unadjuvanted A/H7N9 vaccine, as compared to baseline assessments performed prior to vaccination (Days -7, 1, and 29).

# **Secondary Endpoints**

- 1. Plasma measurement of cytokines and chemokines at each study visit, comparing:
  - a. Post-vaccination time points with pre-vaccination time points by treatment arms.
  - b. AS03-adjuvanted influenza A/H7N9 responses to unadjuvanted influenza A/H7N9 responses.
  - c. Influenza A/H3N2v vaccine to unadjuvanted influenza A/H7N9 vaccine.
  - d. Influenza A/H3N2v vaccine to adjuvanted A/H7N9 vaccine.
- 2. Serologic response to influenza hemagglutinin:
  - a. Percentage of subjects achieving seroconversion (defined as either a pre-vaccination Neut titer <1:10 and a post-vaccination Neut titer ≥1:40 or a pre-vaccination Neut titer ≥1:10 and a minimum four-fold rise in post-vaccination Neut titer) at approximately 28 days after the second study vaccination (A/H7N9 vaccine, with and without adjuvant).

- b. Percentage of subjects achieving seroconversion at approximately 28 days after the study vaccination with influenza A/H3N2v vaccine.
- c. Geometric Mean Titers of serum HAI and Neut antibody at baseline (Day -7 and 1) and 28 days after influenza A/H3N2v vaccination.
- d. Geometric Mean Titers of serum HAI and Neut antibody at baseline (Day -7 and 1), and 28 days after both the first and the second dose of influenza A/H7N9 vaccine (with and without adjuvant).
- 3. Number of differentially expressed genes based on RNA-Seq analysis in human immune cells at Days 2, 4, and 8 after study vaccination, as compared to baseline assessments (Days -7 and 1) after influenza A/H3N2v vaccine.

#### **Tertiary Endpoints**

- 1. Occurrence of solicited local reactogenicity events within 7 days after each study vaccination.
- 2. Occurrence of solicited systemic reactogenicity events within 7 days after each study vaccination.
- 3. Occurrence of unsolicited AEs collected for approximately 28 days after last study vaccination.
- 4. Occurrence of SAEs and MAAEs including new-onset chronic medical conditions and potentially immune-mediated medical conditions for approximately 1 month (A/H3N2v arm) and 12 months (A/H7N9 arms) after last study vaccination.
- 5. Number of differentially abundant proteins based on protein abundance as determined by quantitative proteomics in human immune cells at Days 2, 4, and 8 after study vaccination, as compared to baseline assessments (Days -7 and 1) after influenza A/H3N2v vaccine.
- 6. Number of differentially abundant proteins based on protein abundance as determined by quantitative proteomics analysis, in human immune cells at Days 2, 4, 29, 30, 32, and 36 after study vaccination with AS03-adjuvanted and unadjuvanted A/H7N9 vaccine comparing changes in protein abundance between treatment arms (A/H7N9 vaccine vs. A/H7N9 vaccine + AS03).

#### **Exploratory Endpoints**

- 1. RNA expression, clusters of co-expressed genes, enriched pathways, and other functional modules as determined by RNA-Seq analysis, in human immune cells at Days 2, 4, 29, 30, 32, and 36 after study vaccination with AS03-adjuvanted and unadjuvanted A/H7N9 vaccine comparing changes in RNA expression between treatment arms (A/H7N9 vaccine vs. A/H7N9 vaccine + AS03).
- 2. Protein abundance, clusters of co-abundant proteins, enriched pathways, and other functional modules as determined by quantitative proteomics analysis, in human immune cells at Days 2, 4, 29, 30, 32, and 36 after study vaccination with AS03-adjuvanted and unadjuvanted A/H7N9 vaccine comparing changes in protein abundance between treatment arms (A/H7N9 vaccine vs. A/H7N9 vaccine + AS03).
- 3. RNA expression, clusters of co-expressed genes, enriched pathways, and other functional modules as determined by RNA-Seq analysis, in human immune cells at Days 2, 4, and 29 after study vaccination comparing baseline changes in RNA expression between treatment arms (A/H3N2v vaccine vs. A/H7N9 vaccine and A/H3N2v vaccine vs. A/H7N9 vaccine + AS03).
- 4. Protein abundance, clusters of co-abundant proteins, enriched pathways, and other functional modules as determined by quantitative proteomics analysis, in human immune cells at Days 2, 4, and 29 after first study vaccination comparing baseline changes (Days -7, and 1) in protein abundance between

- treatment arms (A/H3N2v vaccine vs. A/H7N9 vaccine and A/H3N2v vaccine vs. A/H7N9 vaccine + AS03).
- 5. Changes from baseline (Days -7, 1, and 29) in RNA expression or protein abundance that best correlate with influenza A/H7N9 seroconversion and with peak HAI titers at Days 2 and 4 (following first study vaccination) as well as Days 30, 32, and 36 (following second study vaccination).
- 6. Changes from baseline (Days -7, 1, and 29) in RNA expression or protein abundance that best correlate with baseline changes in cytokine concentrations at Days 2, 4, 8 (A/H3N2v arm only) and 29 (following first study vaccination) as well as Days 30, 32, and 36 (following second study vaccination).
- 7. Exploratory summaries of transcriptomics/proteomics response signatures for subjects with unexpected or severe safety profiles.
- 8. Lists of differential genes and proteins identified as part of the primary and secondary objectives.

# 3.3. Study Definitions and Derived Variables

Derived safety variables are described in Table 3, Table 4, Table 5, Table 6, and Table 7 in this document. The following assay-specific criteria will be used to determine seroconversion for the hemagglutination inhibition (HAI) and neutralization (NT) titers:

• a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and a minimum of a four-fold rise in post-vaccination antibody titer.

# 4. INVESTIGATIONAL PLAN

# 4.1. Overall Study Design and Plan

This is a single center, randomized, partially-blinded, Phase II, small, targeted, prospective study in approximately 30 healthy male and non-pregnant female subjects aged 18 to 49 years old, inclusive, designed to evaluate and compare the immunogenicity between an intramuscular monovalent inactivated influenza A/H7N9 virus vaccine manufactured by Sanofi Pasteur given with and without AS03 adjuvant manufactured by GlaxoSmithKline, and an intramuscular unadjuvanted monovalent inactivated influenza A/H3N2v virus vaccine manufactured by Sanofi Pasteur.

This study will use a standard and systems biology approach to assess the human early gene and protein signatures expressed at baseline (approximately Days -7 and 1), and at approximately Days 2, 4, and 8 (A/H3N2v-vaccinated subjects only) after the first study vaccination in each treatment arm as well as at approximately Days 29, 30, 32, and 36 in A/H7N9-vaccinated subjects only. Cellular immunogenicity (systems biology studies) data will be integrated with serologic immunogenicity (HAI and Neut antibody assays) and reactogenicity data to develop a systems model of the human immune response to unadjuvanted monovalent inactivated influenza A/H3N2v virus vaccine and monovalent inactivated influenza A/H7N9 virus vaccine given with and without ASO3 adjuvant.

This study will use venous blood samples and subject data collected from a total of thirty vaccinated subjects randomly divided into three equal treatment arms (Table 1). The first treatment arm (n=10) will be vaccinated with one dose of 15  $\mu$ g of A/H3N2v HA. The second treatment arm (n=10) will be vaccinated with two doses of 3.75  $\mu$ g of A/H7N9 HA given with AS03 approximately 28 days apart. The third treatment arm (n=10) will be vaccinated with two doses of 3.75  $\mu$ g of A/H7N9 HA given without AS03 adjuvant approximately 28 days apart. All study vaccinations will be administered intramuscularly.

Reactogenicity will be measured by the occurrence of solicited injection site and systemic reactions from the time of each study vaccination through 8 days after each study vaccination. Unsolicited non-serious adverse events (AEs) will be collected from the time of each study vaccination through approximately 28 days after each study vaccination. Serious adverse events (SAEs) and medically-attended adverse events (MAAEs) including new-onset chronic medical conditions (NOCMCs) and potentially immune-mediated medical conditions (PIMMCs) will be collected from the time of the first study vaccination through approximately 1 month (A/H3N2v arm) and 12 months (A/H7N9 arms) after the last study vaccination.

Venous blood samples (approximately 90 mL) will be collected from subjects at approximately Days -7 and 1 (immediately prior to the first study vaccination), and at approximately Days 2, 4; and 8 (A/H3N2v-vaccinated subjects only) after the first study vaccination for systems biology studies (cytokine and chemokine levels, immune cell activation status, and whole transcriptome and proteome profiles of the major blood immune cells). Additionally, subjects in either treatment arm receiving A/H7N9 vaccine will have additional blood samples collected at approximately Days 29 (this will be collected immediately prior to the second study vaccination for subjects in either group receiving A/H7N9), 30, 32, and 36 after the first study vaccination for systems biology studies.

Serological assessment (hemagglutination inhibition (HAI) and neutralizing (Neut) antibody assays) will also be conducted on venous blood samples (approximately 10 mL) collected from subjects at Day 1 (immediately prior to the first study vaccination), and at approximately Days 29 (for A/H7N9-vaccinated subjects this will be collected immediately prior to the second study vaccination) and 57 (A/H7N9-vaccinated subjects only) after the first study vaccination. Plasma cytokine/chemokine levels, as well as transcriptomic and proteomic

profiles from individual immune cell compartments will be measured and integrated with standard serologic assessment to vaccine.

Urine samples (approximately 20 mL) will also be collected from subjects at approximately Days -7, 1, 2, 4, 8 (A/H3N2v-vaccinated subjects only), 29, 30, 32, and 36 for future research.

# 4.2. Discussion of Study Design, Including the Choice of Control Groups

The main study arms are the two arms receiving influenza A/H7N9 virus vaccine with or without AS03 adjuvant (Study Arms 2 and 3). The goal is to better understand how the AS03 adjuvant modulates the immune response to influenza A/H7N9 virus on the molecular level. The addition of the interpandemic (seasonal) strain of influenza A/H3N2v was chosen to compare innate and adaptive immune response between avian (A/H7N9) and swine-origin influenza vaccines (A/H3N2v) more closely resembling seasonal strains of influenza A.

# 4.3. Selection of Study Population

#### **Subject Inclusion Criteria**

Subjects eligible to participate in this study must meet all of the following inclusion criteria:

- 1. Provide written informed consent prior to initiation of any study procedures.
- 2. Are able to understand and comply with planned study procedures and be available for all study visits.
- 3. Are males or non-pregnant females, 18 to 49 years old, inclusive.
- 4. Are in good health<sup>1</sup>.

<sup>1</sup>As determined by medical history and targeted physical examination, if indicated based on medical history, to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days, that would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days. This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change, and there is no additional risk to the subject or interference with the evaluation of responses to study vaccination. Note: Topical, nasal, and inhaled medications (with the exception of inhaled corticosteroids as outlined in the Subject Exclusion Criteria (see Section 5.1.2)), herbals, vitamins, and supplements are permitted.

- 5. Oral temperature is less than 100.4°F.
- 6. Pulse is 50 to 115 bpm, inclusive.
- 7. Systolic blood pressure is 85 to 150 mm Hg, inclusive.
- 8. Diastolic blood pressure is 55 to 95 mm Hg, inclusive.
- 9. Erythrocyte sedimentation rate (ESR) is less than 30 mm per hour.

10. Women of childbearing potential<sup>2</sup> must use an acceptable contraception method<sup>3</sup> from 30 days before first study vaccination until 60 days after last study vaccination.

11. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study vaccination.

# **Subject Exclusion Criteria**

Subjects eligible to participate in this study must not meet any of the following exclusion criteria:

1. Have an acute illness<sup>4</sup>, as determined by the site principal investigator or appropriate sub-investigator, within 72 hours prior to study vaccination.

<sup>4</sup>An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site principal investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.

2. Have any medical disease or condition that, in the opinion of the site principal investigator or appropriate sub-investigator, is a contraindication to study participation<sup>5</sup>.

<sup>5</sup>Including acute or chronic medical disease or condition, defined as persisting for at least 90 days that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this study.

- 3. Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
- 4. Have known active neoplastic disease (excluding non-melanoma skin cancer) or a history of any hematologic malignancy.
- 5. Have known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection.
- 6. Have known hypersensitivity or allergy to eggs, egg or chicken protein, squalene-based adjuvants, or other components of the study vaccines.
- 7. Have a history of severe reactions following previous immunization with licensed or unlicensed influenza virus vaccines.
- 8. Have a personal or family history of narcolepsy.
- 9. Have a history of Guillain-Barré syndrome.
- 10. Have a history of convulsions or encephalomyelitis within 90 days prior to study vaccination.

 $<sup>^2</sup>$ Not sterilized via tubal ligation, bilateral oophorectomy, hysterectomy or successful Essure<sup>®</sup> placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year of the last menses if menopausal.

<sup>&</sup>lt;sup>3</sup>Includes, but is not limited to, non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving the first study vaccination, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing<sup>®</sup>, and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill").

11. Have a history of a potentially immune-mediated medical condition<sup>6</sup>.

<sup>6</sup>Refer to Appendix A: List of Potentially Immune-Mediated Medical Conditions.

- 12. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
- 13. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
- 14. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
- 15. Have taken oral or parenteral (including intra-articular) corticosteroids of any dose within 30 days prior to study vaccination.
- 16. Have taken high-dose inhaled corticosteroids within 30 days prior to study vaccination. High-dose defined as >840 mcg/day of beclomethasone dipropionate CFC or equivalent.
- 17. Received licensed live vaccine within 30 days prior to the first study vaccination, or plans to receive licensed live vaccine within 30 days before or after each study vaccination.
- 18. Received licensed inactivated vaccine within 14 days prior to the first study vaccination, or plans to receive licensed inactivated vaccine within 14 days before or after each study vaccination.
- 19. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 90 days prior to study vaccination.
- 20. Received an experimental agent<sup>7</sup> within 30 days prior to the first study vaccination, or expects to receive an experimental agent<sup>8</sup> during the 13-month study-reporting period.

<sup>7</sup>Including vaccine, drug, biologic, device, blood product, or medication.

<sup>8</sup>Other than from participation in this study.

21. Are participating or plan to participate in another clinical trial with an interventional agent<sup>9</sup> that will be received during the 13-month study-reporting period.

<sup>9</sup>Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.

22. Prior participation in a clinical trial of influenza A/H7 vaccine<sup>10</sup> or have a history of influenza A/H7 virus actual or potential exposure or infection prior to the first study vaccination.

<sup>10</sup>And assigned to a group receiving influenza A/H7 vaccine, does not apply to documented placebo recipients.

23. Prior participation in a clinical trial of influenza A/H3N2v vaccine<sup>11</sup> or have a history of influenza A/H3N2v virus actual or potential exposure or infection prior to the first study vaccination.

<sup>11</sup>And assigned to a group receiving influenza A/H3N2v vaccine, does not apply to documented placebo recipients.

24. Occupational exposure to or substantial direct physical contact<sup>12</sup> with birds in the past year or during the 28 days after each study vaccination.

<sup>12</sup>Casual contact with birds at petting zoos or county or state fairs or having pet birds does not exclude subjects from study participation.

25. Occupational exposure to or substantial direct physical contact<sup>13</sup> with pigs in the past year or during the 28 days after each study vaccination.

<sup>13</sup>Casual contact with pigs at petting zoos or county or state fairs does not exclude subjects from study participation.

- 26. Female subjects who are breastfeeding or plan to breastfeed at any given time from the first study vaccination until 30 days after the last study vaccination.
- 27. Plan to travel outside the US (continental US, Hawaii, and Alaska) within 28 days after each study vaccination.
- 28. Blood donation or planned blood donation within 30 days before enrollment until 30 days after the last blood draw for this study.

#### 4.4. Treatments

#### 4.4.1. Treatments Administered

#### A/H7N9 Vaccine

Sanofi Pasteur has developed a monovalent inactivated influenza A/H7N9 virus vaccine for intramuscular use. The manufacturing process for the production of this monovalent inactivated influenza A/H7N9 virus vaccine is similar to the manufacturing process for the production of its licensed Influenza Virus Vaccine Fluzone® family of products, except for a minor modification in the PBS diluent in the formulation step that was made according to previous experiences of manufacturing of monovalent pandemic vaccines. This monovalent inactivated split influenza virus vaccine was derived from the influenza A/Shanghai/2/2013 virus. Licensed release testing specifications were maintained, with a modification to the potency test.

A 3.75 mcg of HA (A/Shanghai/2/2013) per 0.5 mL [adjuvanted] or 0.25 mL [unadjuvanted] dose was planned for use in this study.

AS03 Adjuvant [Adjuvant System (03)]

#### A/H3N2v Vaccine

Sanofi Pasteur has developed a monovalent inactivated influenza A/H3N2v. The resulting reassortant is designated A/Minnesota/11/2010 NYMC X-203 virus vaccine for intramuscular use. The manufacturing process for the production of this monovalent inactivated influenza A/H3N2v virus vaccine is similar, with

slight modifications in the formulation step, to the manufacturing process for the production of its licensed Influenza Virus Vaccine Fluzone® and the H1N1 influenza vaccine A/California/07/2009 NYMC X-179A. Using the Fluzone® production process, an A/H3N2v reassortant was derived from the A/Minnesota/11/2010 strain produced by classical reassortant technology at New York Medical College (NYMC) and provided by the Centers for Disease Control and Prevention (CDC). This monovalent inactivated split influenza virus vaccine is prepared from influenza virus propagated in embryonated chicken eggs. Licensed release testing specifications were maintained

#### 4.4.2. Identity of Investigational Product(s)

#### A/H7N9 Vaccine

The monovalent inactivated influenza A/H7N9 virus vaccine was supplied as a sterile, clear, and slightly opalescent suspension in single-dose vials containing 7.5 mcg of HA per 0.5 mL. Each vial contained a fill volume of 0.7 mL. It contained no preservative (i.e., non-thimerosal) or antibiotics. The vials containing study product had to be stored at 2°C to 8°C (35.6°F to 46.4°F) and not frozen. Vials were provided with latex-free stoppers.

#### AS03 Adjuvant

The AS03 adjuvant was supplied as a preservative-free, oil-in-water, whitish to yellowish homogenous milky liquid emulsion in single-use vials containing a fill volume of 3.15 mL. The vials containing study product had to be stored at 2°C to 8°C (35.6°F to 46.4°F) and not frozen. Vials were provided with latex-free stoppers.

#### A/H3N2v Vaccine

The monovalent inactivated influenza A/H3N2v virus vaccine was supplied as a sterile, clear, and slightly opalescent suspension. A minor modification in the PBS diluent in the formulation step was made to accommodate the nature of the diluted virus in single-dose, prefilled syringes, without needles, containing 15 mcg of HA per 0.5mL. It contained no preservative (i.e., non-thimerosal), antibiotics, or latex. The vaccine included porcine gelatin (0.05%) as a stabilizer. The prefilled syringes containing study product had to be stored at 2°C to 8°C (35°F to 46°F) and not frozen.

Each of these study products were labeled according to manufacturer specifications and included the statement "Caution: New Drug – Limited by Federal Law to Investigational Use."

Further details are included in the respective, applicable Investigator's Brochures and Supplemental Information for the Investigator's Brochures for the A/H7N9 vaccine, AS03 adjuvant, and A/H3N2v vaccine as well as protocol-specific MOP.

#### 4.4.3. Method of Assigning Subjects to Treatment Groups (Randomization)

Per International Conference on Harmonisation (ICH) guideline E6: Good Clinical Practice (GCP), screening records were kept at the participating VTEU site to document the reason why an individual was screened, but failed study entry criteria. The reasons why individuals failed screening were recorded in the Statistical and Data Coordinating Center's (SDCC) AdvantageEDC<sup>SM</sup> (Electronic Data Capture System).

Once consented and upon entry of demographic data and confirmation of eligibility for this study, the subject was enrolled. Subjects were assigned randomly to 1 of 3 treatment arms (Table 1). The first treatment arm (n=10) was vaccinated with one dose of 15  $\mu$ g of A/H3N2v HA. The second treatment arm (n=10) was vaccinated with two doses of 3.75  $\mu$ g of A/H7N9 HA given with ASO3 approximately 28 days apart. The

third treatment arm (n=10) was vaccinated with two doses of 3.75 µg of A/H7N9 HA given without AS03 adjuvant approximately 28 days apart. All study vaccinations were administered intramuscularly.

Enrollment of subjects was done online using the enrollment module of AdvantageEDC<sup>SM</sup>. The randomization code was prepared by statisticians at the SDCC and included in the enrollment module for this study. AdvantageEDC<sup>SM</sup> assigned each subject to a treatment arm after the demographic and eligibility data had been entered into the system. A designated individual at the participating VTEU site was provided with a code list for emergency unblinding purposes, which was to be kept in a secure place.

# 4.4.4. Selection of Doses in the Study

As with other avian influenza strains, the immunogenicity of inactivated vaccines is poor. Higher doses of hemagglutinin (HA), a major target of the protective immune response, has been shown to generate more frequent and higher antibody titers. Thus, two doses of 3.75 mcg of HA (A/Shanghai/2/2013) were administered for the A/H7N9 arms. Standard dosing of 15 mcg of HA (A/H3N2v) was chosen to more closely resemble the dosing administered as part of seasonal influenza vaccination. While 15 mcg represents a 4-fold increase in HA amount, the vaccine was unadjuvanted and matches what is formulated in seasonal standard dose inactivated influenza vaccines.

# 4.4.5. Selection and Timing of Dose for Each Subject

The dose of vaccine was chosen primarily to mirror the amount provided in DMID 10-0074 in which 3.75 mcg of influenza A/H5N1 virus vaccine was given with or without AS03. This reduced amount represents the minimal amount of HA needed to generate an immune response in the presence of an oil-in-water adjuvant system, based on prior studies. The HA content was kept the same for the unadjuvanted dose in an effort to measure the adjuvant effect specifically. Further, in previous studies, two doses of avian-strain influenza vaccine were required to generate an adaptive response, and typically the second dose was given 3-4 weeks after the first dose.

#### 4.4.6. Blinding

This was a partially-blind clinical study as the unadjuvanted A/H3N2v vaccine treatment arm was open-label to avoid the need for placebo administration at approximately Day 29. Investigators and study personnel remained blinded to allocation of A/H7N9 with or without AS03. The randomization scheme was generated by the SDCC and provided to unblinded study personnel (i.e., research pharmacists performing study vaccination preparations and unblinded study vaccine administrators) at the participating VTEU site. The unblinded study vaccine administrator was a study personnel member credentialed to administer vaccines and may also have participated in dose preparation but was not involved in study-related assessments or had subject contact for data collection following study vaccine administration.

# 4.4.7. Prior and Concomitant Therapy

Administration of any medications, therapies, or vaccines was recorded on the appropriate data collection form. Concomitant medications included all current medications and medications taken within 60 days prior to signing the informed consent form through approximately 28 days after the last study vaccination or through the early termination visit (if prior to 28 days after the last study vaccination), whichever occurred first. Medications reported in the electronic case report form (eCRF) were limited to those taken within 30 days prior to the first study vaccination through approximately 28 days after the last study vaccination. Prescription and over-the-counter drugs were included as well as herbals, vitamins and supplements. In addition, receipt of non-study influenza vaccines was solicited through approximately 28 days after the last

study vaccination and reported in the eCRF. Use of new medication should have prompted evaluation for the presence of a new diagnosis of chronic medical disease or condition. Medications that might interfere with the evaluation of the investigational product(s) should not be have been used during the study-reporting period (approximately 12 months after the last study vaccination) unless clinically indicated as part of the subject's health care. Medications in this category included the prohibited medications per the Subject Exclusion Criteria (see Section 4.3). In addition, the site principal investigator or appropriate sub-investigator may identify other medications that should not have been used due to a risk to subject safety or assessment of reactogenicity and immunogenicity.

#### 4.4.8. Treatment Compliance

Study product was administered to subjects by an unblinded study vaccine administrator via intramuscular (IM) injection at all dosing times according to subject treatment assignment and as described in Section 6.2 in the protocol. The number of administered vaccine doses was recorded.

# 4.5. Immunogenicity and Safety Variables

The following section describes the collection of safety and immunogenicity variables. For a detailed schedule of activities refer to Appendix B of the protocol.

# 4.5.1. Immunogenicity Variables

Venous blood samples (approximately 10 mL) for HAI and Neut antibody assays were collected from subjects at Day 1 (immediately prior to the first study vaccination), and at approximately Days 29 (for A/H7N9-vaccinated subjects this was collected immediately prior to the second study vaccination) and 57 (A/H7N9-vaccinated subjects only) after the first study vaccination. Subjects who withdrew early had HAI and Neut antibody assays run on available sera, including sera from the early termination visit, if available.

Individual HAI and Neut results will be reported by the central immunology laboratory for the A/Shanghai/02/2013xPR8 vaccine strain and the A/Minnesota/11/2010 vaccine strain for the A/H3N2v study arm. Assay results will be reported as a reciprocal titer with values of  $10*2^k$ , where k=0, 1, 2, etc. The lower limit of detection for the HAI and Neut assays is 1:10; values below the limit of detection will be imputed for analysis using one-half the limit of detection (10/2 = 5). For analysis, the geometric mean (calculated on natural log scale) of repeated results for each sample will be computed and used as the response for all subsequent calculations. The variation arising from multiple measurements for an individual at a single time point will not be used in subsequent calculations/statistics. See Section 3.3 for definitions of derived variables for the analysis of HAI and Neut data.

Cytokine and chemokine levels in plasma obtained from venous blood samples were quantitatively measured at approximately Days -7, 1, 2, 4, and 8 (A/H3N2v-vaccinated subjects only) and at approximately Days 29, 30, 32, and 36 for A/H7N9-vaccinated subjects only using the Luminex platform. Cytokine and chemokine levels will be reported as concentrations. Values below the plate-specific LOD for each cytokine and chemokine will be imputed using 1/2 LOD.

#### 4.5.2. -Omics Variables

Transcriptome profiling using RNA-Seq was performed on immune cell subsets collected at approximately Days -7, 1, 2, 4, and 8 (A/H3N2v-vaccinated subjects only) and at approximately Days 29, 30, 32, and 36 for A/H7N9-vaccinated subjects only. Total RNA was isolated using standard methods and subjected to ultra-

high-throughput parallel next generation sequencing. Gene expression levels for each gene were estimated based on the number of mapping sequencing reads.

Proteomics profiling was based on shotgun proteomics using multidimensional liquid chromatography coupled with tandem mass spectrometry and performed on immune cell samples collected at approximately Days -7, 1, 2, 4, and 8 (A/H3N2v-vaccinated subjects only) and at approximately Days 29, 30, 32, and 36 for A/H7N9-vaccinated subjects only. Protein abundance levels for each protein were estimated based on the sample peak intensity ratio compared to the sample that was prepared using a pool of all samples.

#### 4.5.3. Safety Variables

Safety assessments included:

- 1. Study vaccine-related serious adverse events occurring from the time of the first study vaccination through approximately 1 month (A/H3N2v arm) and 12 months (A/H7N9 arms) after the last study vaccination.
- 2. Solicited Adverse Events reactogenicity events occurring from the time of each study vaccination through 7 days after each study vaccination:
  - a) Injection site reactions including pruritus (itching), ecchymosis (bruising), erythema (redness), induration (hardness)/swelling, pain, and tenderness.
  - b) Systemic reactions including fever, feverishness (chills/shivering/sweating), fatigue (tiredness), malaise (general unwell feeling), myalgia (body aches/muscular pain exclusive of the injection site), arthralgia (joint pain exclusive of the injection site), headache, and nausea.
- 3. Unsolicited Adverse Events study vaccine-related non-serious adverse events occurring from the time of each study vaccination through approximately 28 days after each study vaccination.
- 4. Medically-Attended Adverse Events including new-onset chronic medical conditions and potentially immune-mediated medical conditions occurring from the time of the first study vaccination through approximately 1 month (A/H3N2v arm) and 12 months (A/H7N9 arms) after the last study vaccination.

# 5. SAMPLE SIZE CONSIDERATIONS

The sample size is not based on a formal hypothesis. Rather it is based on practical considerations with the goal of gathering enough information to learn more about immune system responses to the vaccine/adjuvant on the molecular level. DMID Protocol 10-0074, entitled: "A Randomized, Double-Blinded, Controlled, Phase I Study in Healthy Adults to Assess the Safety, Reactogenicity, and Immunogenicity of Intramuscular Subvirion Inactivated Monovalent Influenza A/H5N1 Virus Vaccine Administered With and Without AS03 Adjuvant: Standard & Systems Biology Analyses", showed that sample sizes in this range are sufficient to detect key differential signals and carry out systems biology analyses.

#### 6. GENERAL STATISTICAL CONSIDERATIONS

# **6.1.** General Principles

Continuous variables will be summarized using descriptive statistics (n, mean, standard deviation, median, interquartile range (IQR), minimum, and maximum) unless otherwise specified. The frequency and percentages (based on the analysis population size) of observed levels will be reported for all categorical measures. In general, all data will be listed and sorted by study arm and subject, and when appropriate, by study visit number within subject. All summary tables will be structured with a column for each study arm in the following order: Study Arm 1, Study Arm 2, and Study Arm 3.

# **6.2.** Timing of Analyses

The primary CSR will be completed when all primary and secondary endpoint data are available and the data have been cleaned and locked. Any available data from the long-term, tertiary safety follow-up of applicable subjects may also be included. Additional data from the long-term, tertiary safety follow-up of applicable subjects, exploratory correlation analyses, and data from the proteomics portion of the study will be included in one or more addenda to the CSR.

# 6.3. Analysis Populations

# 6.3.1. Safety Analysis Population

The Safety Analysis population includes all subjects who received at least one dose of study vaccine.

# 6.3.2. Intention-to-Treat Analysis (ITT) Population

The intent-to-treat (ITT) population includes all subjects who received at least one dose of study vaccine and contributed both pre- and at least one post-study vaccination blood samples for serological assessment (HAI or Neut antibody assays) for which valid results were reported.

# 6.3.3. Per protocol (PP) Population

The per protocol (PP) population includes all subjects in the ITT subset with the following exclusions:

- Data from all available visits for subjects found to be ineligible at baseline.
- Data from all visits subsequent to major protocol deviations, such as:
  - Second study vaccination not received,
  - Receipt of non-study licensed live vaccine within 30 days before or after each study vaccination,
  - Receipt of non-study licensed inactivated vaccine within 14 days before or after each study vaccination,
  - Receipt of immunosuppressive therapy (e.g., corticosteroids) within 30 days before or after each study vaccination.
  - Data from any visit that occurs substantially out of window. Substantially out of window is
    defined as any visit that occurred outside of the pre-defined protocol window except for the
    following visits for which windows will be redefined as:

- o Day 36: +4/-4
- o Day 57: +7/-4

#### 6.3.4. The -Omics Analysis Population

The 'omics analysis population for the -omics (transcriptomics and proteomics) endpoint analyses will include all subjects who received at least one study vaccination and contributed at least one pre- and one post-vaccination sample for 'omics testing for which valid results were reported. In addition, the following exclusions will be applied:

- post-second dose samples from subjects in Study Arms 2 and 3 that did not receive second vaccination will be excluded.
- samples that were collected substantially out-of-window will be excluded. Substantially out of window is defined as any visit that occurred outside of the pre-defined protocol window except for the following visits for which windows will be redefined as:
  - o Day 36: +4/-4
  - o Day 57: +7/-4

# 6.4. Covariates and Subgroups

There is no *a priori* plan to adjust the analyses of safety and immunogenicity for covariates or to report results by subgroups.

# 6.5. Missing Data

For proteomics data relative protein abundance values will be imputed using the k-nearest neighbors imputation algorithm as implemented in the *impute* R package (See SAP Addendum A for further details). Otherwise, no imputation will be performed for missing values.

# 6.6. Interim Analyses and Data Monitoring

No interim safety or immunogenicity review was conducted.

# 6.7. Multicenter Studies

This was a single site study.

# 6.8. Multiple Comparisons/Multiplicity

No multiple testing adjustments will be carried out for the safety, immunogenicity, and cytokine/chemokine endpoints. For -omics endpoints, the false-discovery rates (FDR) based on the Benjamini-Hochberg procedure as implemented in the R *p.adjust* function will be used to control the false positive rate among significantly differentially expressed genes, proteins, and enriched pathways.

# 7. STUDY SUBJECTS

# 7.1. Disposition of Subjects

A flowchart presenting the disposition of study subjects, adapted from the CONSORT statement will be included (Figure 1). The flowchart will summarize the number of subjects who were eligible, enrolled and randomized, lost to follow-up, and analyzed, by study arm. Screened subjects who were ineligible for enrollment in the study will be presented by inclusion and exclusion criteria (Table 10). A listing of all subjects that received study product is provided in Listing 1. A listing of subjects who discontinued or terminated early from the study will be tabulated in Listing 2. The disposition of subjects in the study will be tabulated by study arm (Table 8). This table will show the number of subjects who were screened, enrolled and received the first vaccination, received both vaccinations, completed -omics blood draws, completed follow-up, and were included in the per-protocol analysis population. For each analysis population, a summary of excluded subjects by study arm and time point will be presented as shown in Table 9. A tabular listing of all subjects, visits, and observations excluded from certain analysis populations will be provided as specified in Listing 5.

# 7.2. Protocol Deviations

A summary of protocol deviations will be presented by the deviation category, type, and study arm in Table 2. This table will provide both the number of subjects and the number of deviations for each category and study arm. All subject-specific protocol deviations and non-subject-specific protocol deviations will be included in Listing 3 and Listing 4, respectively.

#### 8. IMMUNOGENICITY EVALUATION

# 8.1. Serum Antibody Analysis

All immunogenicity analyses will be conducted for both the ITT and PP analysis populations. For each analysis population (ITT and PP) and serum antibody assay (HAI and Neut), geometric mean titers (GMTs and two-sided 95% confidence interval (CI) based on t-distribution) and percent seroconversion ([n/N (%)] and an exact (Clopper-Pearson) two-sided 95% CI as defined in Section 3.3) will be summarized by study arm and post-vaccination time point (Table 14, Table 15, Table 16, Table 17). GMTs over time will be summarized using time trend plots (Figure 2). Subject-level serum antibody titer responses at Day 29 post-last vaccination for all three study arms will be contrasted using bar plots (Figure 3). Differences between the treatments will be evaluated at Day 29 post-last dose using two-sided t-tests adjusting for unequal variance if necessary using a standard t-test or Welch's t-test (Table 18, Table 19, Table 20, Table 21). The decision on whether to adjust for unequal variance will be based on inspection of variances for the three study arms. Differences in seroconversion rates for Day 29 post-last dose will be assessed using a two-sided Fisher's exact test (Table 22, Table 23, Table 24, Table 25). Data listings of HAI and Neut assay results will be provided in Listing 8 sorted by study group, subject ID, and visit.

# 8.2. Plasma Cytokines/Chemokine Analysis

Pre-first vaccination cytokine/chemokine concentration will be determined using the mean concentrations among pre-vaccination measurements at Day -7 to -1 and Day 1. Cytokine/chemokine concentrations as well as their baseline fold changes will be summarized using minimum, Q1, median, Q3, maximum, and 95% CI of the median (starting with Table 26 and ending with Table 121). The 95% CI of the median concentration and median fold change from baseline will be determined by using the bootstrap method using 1,000 bootstrap replicates and will be visualized using time trend plots (Figure 4) and radar plots (Figure 5). To identify cytokines/chemokines that show a differential response from baseline, a two-sided Wilcoxon signed-rank test will be carried out for each study arm and post-vaccination time point (Table 122, Table 123). Significant differences in fold changes between study arms for shared post-vaccination time points will be evaluated using a Wilcoxon rank-sum test (Table 124, Table 125). Data listings of cytokine/chemokine assay results will be provided as shown in Listing 9 sorted by study group, subject ID, and visit.

#### 9. TRANSCRIPTOMICS EVALUATIONS

The following sections describe the analysis of RNA-Seq endpoint data for the main Clinical Study Report. Analysis will be based on the PP analysis population. To the extent possible, transcriptomics analyses will be implemented using the R statistical programming language [1] and will utilize published R packages such as made available via the Bioconductor online resource [2]. At the start of the analysis, the most-up-to-date Bioconductor version, R statistical software, and other third-party software will be identified and used.

# 9.1. RNA-Seq Data Processing and Qc

#### 9.1.1. Human Reference Genome Alignment and Quality Assessment

The latest version of the human reference genome assembly, gene models, and associated gene and transcript annotation information in the form of a Gene Transfer Format (GTF) file will be obtained from the ENSEMBL database [3]. Reference dataset versions will be documented in the CSR. Adapter sequences and low-quality 5' ending sequences will be removed from raw sequencing reads using the Trimmomatic software [4]. The impact of quality filtering will be assessed using FastQC software [5]. Quality-filtered reads will then be aligned to the reference transcriptome/genome using the latest version of HISAT2 splice-aware sequence aligner [6]. For each sample, the quality of reference alignments will be evaluated using the RSeQC software [7]. Quality measures for each laboratory will be summarized in tabular form, univariate boxplots and multivariate starplots (Figure 6).

# 9.1.2. Gene Expression Quantification and Data Normalization

Gene expression quantification will be carried out on the gene level using the featureCounts function of the Subread software [8]. Reads that overlap with multiple genes or map to multiple genomic locations on the reference genome will be excluded. Known ribosomal, transfer, and mitochondrial RNA genes will be removed from the final read count analysis dataset. In addition, genes located on the X and Y chromosomes will be excluded from the final read count analysis dataset to avoid gender-related biases.

Systematic sample differences in sequencing coverage will be corrected for by calculating scaling factors for each sample using the trimmed mean of M-values (TMM) method [9] as implemented in the edgeR software [10]. TMM-normalized moderated log<sub>2</sub> counts per million (LCPM) for each gene will be calculated using the edgeR software [10]. As part of this step, a sequencing coverage—scaled count of 0.5 reads will be added to each gene to avoid taking the log of zero. LCPM distributions will be visualized using univariate boxplots and cumulative distribution function (CDF) plots before and after TMM-normalization.

#### 9.1.3. Global Outlier and Batch Effect Detection

TMM-normalized LCPM will be standardized (z-score: mean=0, variance=1) and LCPM distributions across samples will be inspected for outliers (potential sample mislabeling, experimental error, etc.) and systematic effects (sample ordering, batch processing, etc.) using hierarchical clustering, multidimensional scaling, and principal component analysis (Figure 7). If outlying samples are discovered, corresponding clinical and laboratory metadata will be inspected for abnormalities. Based on these findings, a decision will be made as to whether the respective RNA-Seq observation should be removed from downstream analyses. The decision will be recorded in the CSR. If a noticeable batch effect is observed, unless an imbalance across vaccine groups is observed, the batch effect may be accounted for by adding a batch blocking factor as part of the negative binomial models (see Section 9.2).

#### 9.1.4. Pre-Vaccination Transcriptomics Activity

The two pre-first vaccination time point RNA-Seq samples (Day -7 to -1 and Day 1) measure the baseline transcriptomics activity for each subject enrolled in this study. For each subject, baseline transcriptomic activity will be represented by averaging results for the two pre-first vaccination samples by using the sum of the read counts for each gene followed by TMM normalization as described in Section 9.1.2. Globally outlying Day -7 to -1 or Day 1 RNA-Seq samples will be excluded (see Section 9.1.3). The combined pre-first vaccination sample will be used as a reference to assess transcriptomics responses at Days 2, 4, 8, or 29 post-first vaccination. The Day 29 time point RNA-Seq sample also measures the pre-second vaccination transcriptomics activity for each subject enrolled in this study. This sample will be used as a reference to assess post-second vaccination responses (Days 2, 4, and 8 post-second vaccination) for subjects that received a second vaccine dose (Study Arms 2 and 3).

# 9.1.5. Log Fold Change Calculations

Log<sub>2</sub> fold changes (LFC) per gene for each subject and post-vaccination day will be calculated by subtracting pre-vaccination LCPM values from the respective post-vaccination day LCPM value. Two sets of LFC will be determined to separately assess post-first and post-second vaccination responses:

- 1. Day 2, 4, 8, or 29 vs. pre-first vaccination (averaged Day -7 to -1 and Day 1 results) LCPM for Study Arms 1, 2, and 3.
- 2. Day 30, 32, and 36 vs. pre-second vaccination (Day 29) LCPM for Study Arms 2 and 3

# 9.1.6. Determination of Cut Offs for Filtering Lowly Expressed Genes

Transcriptome-wide LCPM results will be used to identify a suitable minimum LCPM filter cut off to exclude lowly expressed genes excluding outlying samples. Genes with mean normalized expression levels below X log<sub>2</sub> counts per million across all samples (all study arms and time points) will be considered to be lowly expressed and will be excluded from the differential expression analysis. To determine a suitable cut off value for X, reverse cumulative distribution function (RCDF) plots summarizing the percentage of genes that exceeded a certain LCPM cut off will be plotted on the y-axis (Figure 8). The goal is to choose a cut off that retains between 10,000 and 14,000 genes for differential analysis. A default cut off of 1 count per million will be used if the targeted gene coverage is met. The filtered set will be used as input for down-stream transcriptomics endpoint analysis described in subsequent sections.

# 9.2. Identification of Differentially Expressed Genes

Negative binomial generalized linear models as implemented in the edgeR software [10] will be applied to identify differentially expressed (DE) genes after exclusion of outlying samples and lowly expressed genes. TMM-adjusted total read counts per sample will be included in the models as an offset to account for systematic sample differences. If systematic technical bias is detected and the effect is balanced across study arms, it will be accounted for by including a covariate or factor as part of the negative binomial models.

For all study arms, DE gene analysis will be carried out for each post-first vaccination study day (Day 2, 4, 8 or 29) in relation to pre-first vaccination gene expression levels (Section 9.2.1). For Study Arms 2 and 3, DE gene analysis will be carried out for each post-second vaccination study day (Day 30, 32, and 36) in relation to pre-second vaccination (Day 29) gene expression levels (Section 9.2.2). In addition, differences in DE gene responses between Study Arms will be assessed for all possible pairwise study arm comparisons (Section 9.2.3).

To control for testing multiple genes, the false-discovery rate (FDR) based on the Benjamini-Hochberg procedure [12] as implemented in the p.adjust R function will be applied for each model. In all cases, genes with an absolute fold change (effect size) of  $\geq 1.5$  compared to pre-vaccination or between Study Arms and FDR-adjusted p-value < 0.05 will be considered significantly DE. Depending on observed magnitude of differential expression effects, the pre-specified fold change cut off of 1.5-fold may be revised. The number of DE genes will be tabulated by study arm and time point (Table 126 and Table 127). In addition, DE gene listings that include gene annotations,  $\log_2$  fold change estimates, p-values, FDR-adjusted p-values, likelihood ratio statistic and average LCPMs will be provided for each post-vaccination day (Table 128).

Treatment effects in terms of overall fold changes and FDR-adjusted p-values will be summarized for all genes that passed the low expression cut off using MA plots and Volcano plots (Figure 9). Overlap in DE genes between post-vaccination days and Study Arms will be summarized using UpSet plots as outlined in Figure 10 both in terms of overall numbers and separately for up/down- regulated DE genes.

The following sections describe the negative binomial model parameterization and hypotheses that will be tested.

#### 9.2.1. Identification of DE Genes Compared to Pre-First Vaccination

For each post-first vaccination day and study arm, a negative binomial model will be fit to pre- and post-first vaccination read counts. Each model will include coefficients to estimate subject and pre- vs. post-first vaccination effects. The subject effects for estimating subject-specific pre-first vaccination levels will be added to account for paired samples from the same subject. Effects will be parameterized in the design matrix using dummy variables with one variable for each subject and an additional variable for the vaccination effect. For vaccination effects, the value will be set to 1 for post-first vaccination and 0 for pre-first vaccination observations. For each gene, the statistical significance of the post- vs. pre-vaccination effect will be evaluated using a likelihood ratio testing the following hypothesis on the log<sub>2</sub> scale:

$$H_0$$
:  $\mu_{post-vaccination}$  -  $\mu_{pre-vaccination} = 0$ ,  $H_1$ :  $\mu_{post-vaccination}$  -  $\mu_{pre-vaccination} \neq 0$ 

Genes with an absolute fold change (effect size) of  $\geq$  1.5 compared to pre-first vaccination and FDR-adjusted p-value < 0.05 will be considered to be significantly DE.

#### 9.2.2. Identification of DE Genes Compared to Pre-Second Vaccination

For subjects receiving a second vaccination, for each post-second vaccination day (Day 30, 32, and 36) and study arm (Study Arms 2 and 3), a negative binomial model will be fit to pre- and post-second vaccination read counts across subjects. The model will be parameterized and evaluated as described in Section 9.2.1, except using Day 29 as the pre-vaccination reference.

# 9.2.3. Identification of Genes with Differential Responses Between Study Arms

For each shared post-first vaccination day (Day 1, 2 and pairwise study arm comparison, a negative binomial model will be fit to pre- and post-first vaccination read counts across the respective study arm pair (Study Arms 2 vs. 3, Study Arms 2 vs. 1, Arms 3 vs. 1). Each model will include coefficients to estimate subject and pre- vs. post-first vaccination effects for each of the two study arms that are being compared. For each shared post-first vaccination day, genes that significantly differed in their post vs. pre-first vaccination response between study arms will then be identified using contrasts testing the following hypothesis for study arm pair X and Y:

```
H_0: (\mu_{post\text{-vaccination Study Arm X}} - \mu_{pre\text{-vaccination Study Arm X}}) - (\mu_{post\text{-vaccination Study Arm Y}} - \mu_{pre\text{-vaccination Study Arm Y}}) = 0
H_1: (\mu_{post\text{-vaccination Study Arm X}} - \mu_{pre\text{-vaccination Study Arm Y}}) - (\mu_{post\text{-vaccination Study Arm Y}} - \mu_{pre\text{-vaccination Study Arm Y}}) \neq 0
```

Similarly, for all post-second vaccination timepoints, models will be fit to identify DE genes between Study Arm 2 vs. 3 except using Day 29 as the pre-vaccination reference.

Genes with an absolute fold change difference (effect size) of  $\geq 1.5$  in their response between study arms and FDR-adjusted p-value < 0.05 will be considered significantly DE between Study Arms.

# 9.3. Determination of higher order functional and temporal organization of differentially expressed genes

# 9.3.1. Subject-level Response Heatmaps

Per-subject baseline log<sub>2</sub> fold change patterns for DE genes will be visualized across Study Arms for each post-vaccination day and fold change set (post-first vaccination and post-second vaccination) using heatmaps (Figure 11, left panel). Genes identified as DE for any of the comparisons described in Section 9.2 will be included as part of this analysis. Heatmaps will include subject and gene dendrograms based on uncentered Pearson correlation distance and complete linkage hierarchical clustering.

#### 9.3.2. Identification of Co-Expressed Gene Clusters

Unsupervised multiscale bootstrapping as implemented in the pvclust R package [12] will be carried out to identify robust clusters of genes with correlated log<sub>2</sub> fold change responses for each fold change set (post-first vaccination and post-second vaccination). Bootstrap resampling will be based on uncentered Pearson correlation distances between log<sub>2</sub> fold change responses in combination with complete linkage clustering. Genes identified as DE for any of the comparisons described in Section 9.2 will be included as part of this analysis. Clusters with a bootstrap probability > 0.95 and maximum distance between cluster members of 0.5 (equivalent to minimum uncentered Pearson correlation of 0.5 among all members) will be considered robust gene clusters. Resulting robust gene cluster dendrograms will be visualized (Figure 11, middle panel) and cluster information will be tabulated (Table 129). In addition, mean log<sub>2</sub> fold change for robust gene clusters (mean across all member genes in a cluster) and associated 95% bootstrap CIs (1000 replicates each) will be visualized by study arm across the respective post-vaccination days (Figure 11, right panel).

# 9.3.3. Pathway Enrichment Analysis

Pathway enrichment analysis will be carried out separately for each DE gene set identified (post vs. prevaccination as well as between study arm comparisons) using published pathway information obtained from KEGG [13] (KEGG Pathways), MSigDB [14] (MSigDB Reactome Pathways, MSigDB GO Biological Process, and MSigDB Immunologic Signatures), and Blood Transcription Modules [15]. Pathway enrichment analysis will be conducted using the goseq algorithm [16] to adjust for RNA-Seq-specific gene length bias <sup>1</sup>. Pathways with a FDR-adjusted p-value < 0.05 will be considered significantly enriched. Due to the relatively increased number of pathways in the MSigDB Immunologic Signatures set, a more stringent FDR-adjusted

<sup>1</sup> For RNA-Seq, longer genes tend to obtain higher read counts compared to shorter genes as they occupy a higher proportion of the transcriptome/genome space. As such gene expression based on read counts is not only proportional to the actual expression but a combination of read length and actual expression. This results in greater statistical power for detecting differential genes if they are long and highly expressed. The effect needs to be addressed in gene set enrichment analysis as comparisons are made between sets of genes. Otherwise gene sets that on average contain larger genes will more likely be identified as significantly enriched compared to gene sets with on average smaller genes.

p-value < 0.01 will be used. Pathway enrichment results including gene set annotation, gene set size, number of DE genes in a gene set by up and down-regulation, Jaccard similarity index, p-value, and FDR-adjusted p-value will be listed (Table 130). For enriched KEGG pathways, log<sub>2</sub> fold change from baseline will be overlaid on top of pathway maps and significantly up/and down-regulated genes (DE genes) will be highlighted to facilitate visual interpretation (Figure 12, left panel). Overlap between sets of identified enriched pathways will be summarized using UpSet plots (similar to Figure 10). Gene set enrichment trends across study arms and post-vaccination days will be visualized using heatmaps color-coded by enrichment score (-1 x log<sub>10</sub>(enrichment p-value)) (Figure 12, middle panel) as well as time trend plots of median pathway responses (based on median average log<sub>2</sub> fold changes of all pathway members) and associated 95% bootstrap confidence intervals (CIs) (similar to Figure 11, right panel).

# 9.3.4. Protein-Protein Interactions Network Analysis

To further characterize DE genes, experimentally determined protein-protein interaction networks including known Influenza A-host interactions centered around DE genes will be generated using data from the IntAct database [17]. Networks will be visualized using *Cytoscape* [18] (Figure 12, right panel). This analysis will be performed for DE genes that differed between the H7N9 arms.

#### 10. SAFETY EVALUATIONS

Summaries and analysis of safety data will be presented for the Safety Analysis Population. These include reactogenicity following each study vaccination, unsolicited adverse events, and adverse events of special interest including SAEs/MAAEs, new-onset chronic medical conditions, and potentially immune-mediated medical conditions. The goal of the safety summaries is to provide information to guide the exploratory correlation analysis to identify transcriptomic/proteomic changes that are predictive of certain safety profiles. The exploratory correlation analysis will be described in an addendum to this SAP. The following sections describe planned baseline and safety summaries.

# **10.1.** Demographic and Other Baseline Characteristics

Summaries of age, sex, ethnicity, and race will be presented by study arm and overall for all enrolled subjects (Table 11 and Table 12). Ethnicity will be categorized as Hispanic or Latino, or not Hispanic and not Latino. In accordance with NIH reporting policy, subjects may self-designate as belonging to more than one race or may refuse to identify a race, the latter reflected in the CRF as "No" to each racial option. Individual subject listings will be presented for all demographics (Listing 6); pre-existing medical conditions (Listing 7); and concomitant medications (Listing 15). The number of subjects with pre-existing medical conditions by MedDRA System Organ Class and study arm will we provided as shown in Table 13. Summaries of medications that were started prior to dosing and continuing at the time of dosing will be presented by WHO Drug Level 1 and Level 2 codes and study arm for subjects in the safety population (Table 153). The number of doses of study product administered to subjects will be presented by study arm as part of the subject disposition table (Table 8).

#### **10.2.** Adverse Events

# 10.2.1. Solicited Events and Symptoms

Systemic and upper respiratory (local) solicited adverse events were collected pre-vaccination, and systemic and local solicited adverse events were collected 30 minutes post-vaccination and then daily for 7 days after first vaccination and graded on a scale of 0 (absent), 1 (mild), 2 (moderate) and 3 (severe). The grading scales for solicited systemic and local (administration site) adverse events are provided in Table 3, Table 4, Table 5, and Table 6. The percentage of subjects and associated exact Clopper–Pearson 95% CI reporting at least one solicited adverse event will be summarized for each solicited adverse event, any systemic symptom, any local symptom, and any symptoms (Table 132, Table 133, Table 134). In addition, for each systemic and local event, any systemic event, any local event, and any solicited event, the maximum severity over 7 days after each vaccination will be summarized for the Safety population. For each event the denominator is the number of subjects with non-missing data for the specific event (Table 135, Table 136, Table 137). The number of subjects reporting a solicited adverse event will be summarized for each day post vaccination in a summary table (Table 138, Table 139, Table 140, Table 141, Table 142) and graphically in a bar chart (Figure 13). Solicited adverse events by subject will be presented in Listing 10 and Listing 11.

#### 10.2.2. Unsolicited Adverse Events

When calculating the incidence of unsolicited AEs (i.e., on a per subject basis), each subject will only be counted once at the highest severity and/or relationship, and any repetitions of the same AEs within a subject will be ignored; the denominator will be the total number of subjects in the safety population. The number and percentage and associated 95% CI of subjects reporting at least one unsolicited AE will be summarized by MedDRA system organ class and preferred term (Table 143, Table 144, Table 145). Denominators for

percentages are the number of subjects who received the study vaccination summarized. In addition, a summary of the percentage of subjects by MedDRA system organ class, preferred term, severity, and relationship to study product will be provided (Table 146, Table 147, Table 148). Bar charts of the incidence of non-serious adverse events by severity and MedDRA system organ class will be generated as shown in Figure 14. A listing of all reported AEs by subject sorted by study group, subject ID, and AE Number will be presented as specified in Listing 12.

# 10.3. Deaths, Serious Adverse Events and other Significant Adverse Events

The number and percentage of subjects experiencing adverse events of special interest will be tabulated by study arm as presented in Table 131. The following listings will be presented including Subject ID, AE Description, AE Onset Date/End Date, Last Vaccination Received/Days Post Vaccination, Reason Reported as an SAE, Relationship to Treatment, Alternate Etiology if not Related, Outcome, and Duration of Event (days):

- Deaths and Serious Adverse Events (Table 149)
- Non-Serious, Unsolicited, Moderate or Severe Adverse Events (Table 150)
- Adverse Events of Special Interest (Table 151)

# 10.4. Vital Signs and Physical Evaluations

Vital signs will be tabulated by study arm in Table 152. A listing of vital signs will be presented (Listing 13). Targeted physical examinations will be performed, if indicated, based on a subject's medical history. A listing of physical exam findings will be presented (Listing 14).

# 11. TERTIARY AND EXPLORATORY PROTEOMICS ANALYSES

Analysis of tertiary and exploratory endpoints will be described in separate addenda to this SAP which will be finalized prior to analysis of the proteomics data.

# 12. EXPLORATORY CORRELATION ANALYSES

Correlation analysis between the -omics data (transcriptomics and proteomics) and serum antibody/plasma cytokines as well as correlated with certain safety profiles will be described in separate addenda to this SAP which will be finalized prior to the proteomics data lock.
## 13. REPORTING CONVENTIONS

P-values  $\geq$ 0.0001 and  $\leq$ 0.9999 will be reported to 4 decimal places; p-values less than 0.0001 will be reported as "<0.0001"; p-values greater than 0.9999 will be reported as ">0.9999". The mean, standard deviation, and any other statistics other than quantiles, will be reported to one decimal place greater than the original data. Quantiles, such as median, Q1, Q3, minimum and maximum will use the same number of decimal places as the original data.

#### 14. **REFERENCES**

- 1. Statistical Package, R. "R: A language and environment for statistical computing." *Vienna, Austria: R Foundation for Statistical Computing* (2009).
- 2. Gentleman, Robert C., et al. "Bioconductor: open software development for computational biology and bioinformatics." *Genome biology* 5.10 (2004): R80.
- 3. Hubbard, T., et al. "The Ensembl genome database project." *Nucleic acids research* 30.1 (2002): 38-41.
- 4. Bolger, Anthony M., Marc Lohse, and Bjoern Usadel. "Trimmomatic: a flexible trimmer for Illumina sequence data." *Bioinformatics* 30.15 (2014): 2114-2120.
- 5. http://www.bioinformatics.babraham.ac.uk/projects/fastq
- 6. Kim, Daehwan, Ben Langmead, and Steven L. Salzberg. "HISAT: a fast spliced aligner with low memory requirements." *Nature methods* 12.4 (2015): 357.
- 7. Wang, Liguo, Shengqin Wang, and Wei Li. "RSeQC: quality control of RNA-seq experiments." *Bioinformatics* 28.16 (2012): 2184-2185.
- 8. Liao, Yang, Gordon K. Smyth, and Wei Shi. "featureCounts: an efficient general purpose program for assigning sequence reads to genomic features." *Bioinformatics* 30.7 (2014): 923-930.
- 9. Robinson, Mark D., and Alicia Oshlack. "A scaling normalization method for differential expression analysis of RNA-seq data." Genome Biol 11.3 (2010): R25.
- 10. Robinson, Mark D., Davis J. McCarthy, and Gordon K. Smyth. "edgeR: a Bioconductor package for differential expression analysis of digital gene expression data." Bioinformatics 26.1 (2010): 139-140.
- 11. Benjamini, Yoav, and Yosef Hochberg. "Controlling the false discovery rate: a practical and powerful approach to multiple testing." Journal of the Royal Statistical Society. Series B (Methodological) (1995): 289-300.
- 12. Suzuki, Ryota, and Hidetoshi Shimodaira. "Pvclust: an R package for assessing the uncertainty in hierarchical clustering." Bioinformatics 22.12 (2006): 1540-1542.
- 13. Kanehisa, Minoru, and Susumu Goto. "KEGG: kyoto encyclopedia of genes and genomes." Nucleic acids research 28.1 (2000): 27-30.
- 14. Liberzon, Arthur, et al. "Molecular signatures database (MSigDB) 3.0." Bioinformatics 27.12 (2011): 1739-1740.
- 15. Li, Shuzhao, et al. "Molecular signatures of antibody responses derived from a systems biology study of five human vaccines." Nature immunology 15.2 (2014): 195.
- 16. Young, Matthew D., et al. "Method Gene ontology analysis for RNA-seq: accounting for selection bias." Genome Biol 11 (2010): R14.
- 17. Kerrien, Samuel, et al. "IntAct—open source resource for molecular interaction data." *Nucleic acids research* 35.suppl\_1 (2006): D561-D565.
- 18. Shannon, Paul, et al. "Cytoscape: a software environment for integrated models of biomolecular interaction networks." *Genome research* 13.11 (2003): 2498-2504

# 15. LISTING OF TABLES, FIGURES, AND LISTINGS

Table, figure, and listing shells are presented in Appendices 1, 2, and 3.

# **APPENDICES**

# APPENDIX 1. TABLE MOCK-UPS

# LIST OF TABLES

| Table 1: | Study Design and Sample Size | 43 |
|---|---|---|
| Table 2: | Distribution of Protocol Deviations by Category, Type, and Treatment<br>Group | 44 |
| Table 3: | Local (Injection Site) Reactogenicity Grading | 46 |
| Table 4: | Local (Injection Site) Reactogenicity Measurements | 46 |
| Table 5: | Subjective Systemic Reactogenicity Grading | 46 |
| Table 6: | Quantitative Systemic Reactogenicity Grading | 47 |
| Table 7: | Additional Adverse Event Severity Grading | 47 |
| Table 8: | Subject Disposition by Treatment Group – All Enrolled Subjects | 48 |
| Table 9: | Analysis Populations by Treatment Group and Time Point – All Enrolled Subjects | 49 |
| Table 10: | Ineligibility Summary of Screen Failures | 50 |
| Table 11: | Summary of Categorical Demographic and Baseline Characteristics by Treatment Group - All Enrolled Subjects | 51 |
| Table 12: | Summary of Continuous Demographic and Baseline Characteristics by Treatment Group - All Enrolled Subjects | 52 |
| Table 13: | Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group | 53 |
| Table 14: | Summaries of Hemagglutination Inhibition Antibody Titer by Study Day and Treatment Group in the Intent-to-Treat Population | 54 |
| Table 15: | Summaries of Hemagglutination Inhibition Antibody Titer by Study Day and Treatment Group in the Per-Protocol Population | 54 |
| Table 16: | Summaries of Neutralizing Antibody by Study Day and Treatment Group in the Intent-to-Treat Population | 54 |
| Table 17: | Summaries of Neutralizing Antibody by Study Day and Treatment Group in the Per-Protocol Population | 54 |
| Table 18: | t-Test Results for Comparing Day 29 Post-Last Vaccination Hemagglutination Inhibition Antibody Titer between Treatment Groups in the Intent-to-Treat Population | 55 |
| Table 19: | t-Test Results for Comparing Day 29 Post-Last Vaccination Hemagglutination Inhibition Antibody Titer Between Treatment Groups in the Per-Protocol Population | 55 |
| Table 20: | t-Test Results for Comparing Day 29 Post-Last Vaccination Neutralizing Antibody Titer Between Treatment Groups in the Intent-to-Treat Population | 55 |

| Table 21: | t-Test Results for Comparing Day 29 Post-Last Vaccination Neutralizing Antibody Titer Between Treatment Groups in the Per-Protocol Population | 55 |
|---|---|---|
| Table 22: | Fisher's Exact Test Results for Comparing Day 29 Post-Last Vaccination<br>Seroconversion based on Hemagglutination Inhibition Antibody Titer<br>Between Treatment Groups in the Intent-to-Treat Population | 56 |
| Table 23: | Fisher's Exact Test Results for Comparing Day 29 Post-Last Vaccination<br>Seroconversion based on Hemagglutination Inhibition Antibody Titer<br>Between Treatment Groups in the Per-Protocol Population | 56 |
| Table 24: | Fisher's Exact Test Results for Comparing Day 29 Post-Last Vaccination<br>Seroconversion based on Neutralizing Antibody between Treatment Groups<br>in the Intent-to-Treat Population | 56 |
| Table 25: | Fisher's Exact Test Results for Comparing Day 29 Post-Last Vaccination<br>Seroconversion based on Neutralizing Antibody between Treatment Groups<br>in the Per-Protocol Population | 56 |
| Table 26: | Fractalkine Concentration by Study Visit Day and Treatment Group in the Intent-to-Treat Population | 57 |
| Table 27: | Fractalkine Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 59 |
| Table 28: | GM-CSF Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 59 |
| Table 29: | GM-CSF Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 59 |
| Table 30: | Interferon-gamma Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 59 |
| Table 31: | Interferon-gamma Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 59 |
| Table 32: | Interleukin 1 beta Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 59 |
| Table 33: | Interleukin 1 beta Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 59 |
| Table 34: | Interleukin 2 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 59 |
| Table 35: | Interleukin 2 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 59 |
| Table 36: | Interleukin 4 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 59 |
| Table 37: | Interleukin 4 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | |

| Table 38: | Interleukin 5 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 59 |
|---|---|---|
| Table 39: | Interleukin 5 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 59 |
| Table 40: | Interleukin 6 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 59 |
| Table 41: | Interleukin 6 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 59 |
| Table 42: | Interleukin 7 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 59 |
| Table 43: | Interleukin 7 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 60 |
| Table 44: | Interleukin 8 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 60 |
| Table 45: | Interleukin 8 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 60 |
| Table 46: | Interleukin 10 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 60 |
| Table 47: | Interleukin 10 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 60 |
| Table 48: | Interleukin-12, p70 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 60 |
| Table 49: | Interleukin-12, p70 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 60 |
| Table 50: | Interleukin 13 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 60 |
| Table 51: | Interleukin 13 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 60 |
| Table 52: | IL-17A Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 60 |
| Table 53: | IL-17A Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 60 |
| Table 54: | Interleukin 21 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 60 |
| Table 55: | Interleukin 21 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 60 |
| Table 56: | Interleukin 23 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 60 |

| Table 57: | Interleukin 23 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 60 |
|---|---|---|
| Table 58: | Interferon-inducible T Cell Alpha Chemoattractant Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 60 |
| Table 59: | Interferon-inducible T Cell Alpha Chemoattractant Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 60 |
| Table 60: | Macrophage Inflammatory Protein 1 Alpha Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 60 |
| Table 61: | Macrophage Inflammatory Protein 1 Alpha Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 60 |
| Table 62: | Macrophage Inflammatory Protein-1 Beta Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 61 |
| Table 63: | Macrophage Inflammatory Protein-1 Beta Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 61 |
| Table 64: | Macrophage Inflammatory Protein-3 Alpha Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 61 |
| Table 65: | Macrophage Inflammatory Protein-3 Alpha Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 61 |
| Table 66: | Tumor Necrosis Factor Alpha Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 61 |
| Table 67: | Tumor Necrosis Factor Alpha Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 61 |
| Table 68: | Interferon Gamma-Induced Protein 10 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 61 |
| Table 69: | Interferon Gamma-Induced Protein 10 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 61 |
| Table 70: | Interferon-Alpha Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 61 |
| Table 71: | Interferon-Alpha Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 61 |
| Table 72: | Interferon-Beta Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 61 |
| Table 73: | Interferon-Beta Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population | 61 |
| Table 74: | Fractalkine Fold Change by Study Visit Day and Study Group in the Intent-To-Treat Population | 62 |
| Table 75: | Fractalkine Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 64 |

| Table 76: | GM-CSF Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 64 |
|---|---|---|
| Table 77: | GM-CSF Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 64 |
| Table 78: | Interferon-gamma Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 64 |
| Table 79: | Interferon-gamma Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 64 |
| Table 80: | Interleukin 1 beta Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 64 |
| Table 81: | Interleukin 1 beta Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 64 |
| Table 82: | Interleukin 2 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 64 |
| Table 83: | Interleukin 2 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 64 |
| Table 84: | Interleukin 4 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 64 |
| Table 85: | Interleukin 4 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 64 |
| Table 86: | Interleukin 5 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 64 |
| Table 87: | Interleukin 5 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 64 |
| Table 88: | Interleukin 6 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 64 |
| Table 89: | Interleukin 6 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 64 |
| Table 90: | Interleukin 7 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 64 |
| Table 91: | Interleukin 7 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 64 |
| Table 92: | Interleukin 8 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 64 |
| Table 93: | Interleukin 8 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 64 |
| Table 94: | Interleukin 10 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 64 |

| Table 95: | Interleukin 10 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 64 |
|---|---|---|
| Table 96: | Interleukin-12, p70 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 64 |
| Table 97: | Interleukin-12, p70 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 64 |
| Table 98: | Interleukin 13 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 65 |
| Table 99: | Interleukin 13 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 65 |
| Table 100: | IL-17A Fold Change by Study Visit Day and Treatment Group in the Intent-<br>To-Treat Population | 65 |
| Table 101: | IL-17A Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 65 |
| Table 102: | Interleukin 21 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 65 |
| Table 103: | Interleukin 21 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 65 |
| Table 104: | Interleukin 23 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 65 |
| Table 105: | Interleukin 23 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 65 |
| Table 106: | Interferon-inducible T Cell Alpha Chemoattractant Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 65 |
| Table 107: | Interferon-inducible T Cell Alpha Chemoattractant Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 65 |
| Table 108: | Macrophage Inflammatory Protein 1 Alpha Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | |
| Table 109: | Macrophage Inflammatory Protein 1 Alpha Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 65 |
| Table 110: | Macrophage Inflammatory Protein-1 Beta Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | |
| Table 111: | Macrophage Inflammatory Protein-1 Beta Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | |
| Table 112: | Macrophage Inflammatory Protein-3 Alpha Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | |
| Table 113: | Macrophage Inflammatory Protein-3 Alpha Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | |

| Table 114: | Tumor Necrosis Factor Alpha Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | .65 |
|---|---|---|
| Table 115: | Tumor Necrosis Factor Alpha Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | .65 |
| Table 116: | Interferon Gamma-Induced Protein 10 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 65 |
| Table 117: | Interferon Gamma-Induced Protein 10 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 66 |
| Table 118: | Interferon-Alpha Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 66 |
| Table 119: | Interferon-Alpha Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 66 |
| Table 120: | Interferon-Beta Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population | 66 |
| Table 121: | Interferon-Beta Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population | 66 |
| Table 122: | Wilcoxon Signed-Rank Test Results for Comparing Cytokine/Chemokine Concentrations between Pre- and Post-Vaccination Time Points in the Intent-To-Treat Population | .67 |
| Table 123: | Wilcoxon Signed-Rank Test Results for Comparing Cytokine/Chemokine<br>Concentrations between Pre- and Post-Vaccination Time Points in the Per-<br>Protocol Population | .68 |
| Table 124: | Wilcoxon Rank Sum Test Results for Comparing Fold Changes between Study Groups in the Intent-To-Treat Population | |
| Table 125: | Wilcoxon Rank Sum Test Results for Comparing Fold Changes between Study Groups in the Per-Protocol Population | .70 |
| Table 126: | Genes Differentially Expressed Compared to Pre-Vaccination by Treatment Group, Cell Type, and Post-Vaccination Day | 71 |
| Table 127: | Genes Differentially Expressed Between Treatment Groups by Immune Cell Type, and Post-Vaccination Day | .73 |
| Table 128: | Genes Differentially Expressed at Day 2 Compared to Pre-First Vaccination (RNA-Seq, Monocytes, Study Arm 1 A/H3N2v, D1) | .75 |
| Table 129: | Clusters of Co-Expressed Differential Genes (Monocytes, Days 2-29) | 76 |
| | KEGG Pathways Enriched in Differentially Expressed Genes at Day 2<br>Compared to Pre-First Vaccination (RNA-Seq, Monocytes, Study Arm 1<br>A/H3N2v, D1) | |
| Table 131: | Number and Percentage of Subjects Experiencing Adverse Events of Special Interest | |

| Table 132: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, and Treatment Group (Post-First Vaccination) | 79 |
|---|---|---|
| Table 133: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, and Treatment Group (Post-Second Vaccination) | |
| Table 134: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, and Treatment Group (Post-Any Vaccination) | 79 |
| Table 135: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group (Post-First Vaccination) | 80 |
| Table 136: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group (Post-Second Vaccination) | 81 |
| Table 137: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group (Post-Any Vaccination) | 81 |
| Table 138: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Post-Vaccination Day (Post-First Vaccination, Study Arm 1 A/H3N2v, D1) | |
| Table 139: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Post-Vaccination Day (Post-First Vaccination, Study Arm 2 A/H7N9 + AS03, D1, 29) | |
| Table 140: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Post-Vaccination Day (Post-First Vaccination, Study Arm 3 A/H7N9 + PBS, D1, 29) | |
| Table 141: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Post-Vaccination Day (Post-Second Vaccination, Study Arm 2 A/H7N9 + AS03, D1, D29) | |
| Table 142: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Post-Vaccination Day (Post-Second Vaccination, Study Arm 3 A/H7N9 + PBS, D1, 29) | |
| Table 143: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA® System Organ Class and Preferred Term, and Treatment Group (Post-First Vaccination) | |
| Table 144: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA® System Organ Class and Preferred Term, and Treatment Group (Post-Second Vaccination) | |

| Table 145: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA® System Organ Class and Preferred Term, and Treatment Group (Post-Any Vaccination) | 85 |
|---|---|---|
| Table 146: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Maximum Severity, and Relationship (Study Arm 1 A/H3N2v, D1) | 86 |
| Table 147: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Maximum Severity, Relationship (Study Arm 2 A/H7N9 + AS03, D1, 29) | 86 |
| Table 148: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Maximum Severity, Relationship (Study Arm 3 A/H7N9 + PBS, D1, 29) | 86 |
| Table 149: | Listing of Serious Adverse Events | 87 |
| Table 150: | Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events | 87 |
| Table 151: | Listing of Adverse Events of Special Interest | 88 |
| Table 152: | Vital Signs by Assessment, Maximum Severity, Study Day, and Treatment<br>Group – Any Assessment | 89 |
| Table 153: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group | 91 |

# 9.1 Overall Study Design and Plan Description

**Table 1:** Study Design and Sample Size

| Subjects | First Study Vaccination (Day 1) | Second Study Vaccination<br>(Day 29±2 days) | Study Arm Label |
|---|---|---|---|
| 10 | 15 μg A/H3N2v* | N/A | Study Arm 1<br>A/H3N2v, D1 |
| 10 | 3.75 μg A/H7N9 + AS03 | 3.75 μg A/H7N9 + AS03 | Study Arm 2<br>A/H7N9 + AS03<br>D1, 29 |
| 10 | 3.75 μg A/H7N9+PBS | 3.75 μg A/H7N9 + PBS | Study Arm 3<br>A/H7N9 + PBS, D1, 29 |
| | Total N=30 va | ccinated subjects | |

<sup>\*</sup>Unadjuvanted

# **10.2** Protocol Deviations

Table 2: Distribution of Protocol Deviations by Category, Type, and Treatment Group

| Category | Deviation Type | Study Arm 1<br>A/H3N2v, D1<br>(N=X) | | Study Arm 2<br>A/H7N9 + AS03,<br>D1, 29 (N=X) | | Study Arm 3<br>A/H7N9 + PBS, D1,<br>29 (N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|
| | | No.<br>of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No.<br>of<br>Dev. |
| Eligibility/enrollment | Any type | | | | | | | | |
| | Did not meet inclusion criterion | Х | х | | | x | X | x | x |
| | Met exclusion criterion | | | | | | | | |
| | ICF not signed prior to study procedures | | | | | | | | |
| | Other | | | | | | | | |
| Treatment administration schedule | Any type | | | | | | | | |
| | Out of window visit | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | |
| | Missed treatment administration | | | | | | | | |
| | Delayed treatment administration | | | | | | | | |
| | Other | | | | | | | | |
| Follow-up visit schedule | Any type | | | | | | | | |
| | Out of window visit | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | |
| | Other | | | | | | | | |
| Protocol procedure/assessment | Any type | | | | | | | | |
| | Incorrect version of ICF signed | | | | | | | | |
| | Blood not collected | | | | | | | | |
| | Urine not collected | | | | | | | | |
| | Other specimen not collected | | | | | | | | |
| | Too few aliquots obtained | | | | | | | | |
| | Specimen result not obtained | | | | | | | | |
| | Required procedure not conducted | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | |
| | Study product temperature excursion | | | | | | | | |

Table 2: Distribution of Protocol Deviations by Category, Type, and Treatment Group (continued)

| Category | Deviation Type | A/H3N | Arm 1<br>N2v, D1<br>=X) | Study Arm 2<br>A/H7N9 + AS03,<br>D1, 29 (N=X) | | Study Arm 3<br>A/H7N9 + PBS, D1,<br>29 (N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|
| | | No.<br>of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No.<br>of<br>Dev. |
| | Specimen temperature excursion | | | | | | | | |
| | Other | | | | | | | | |
| Treatment administration | Any type | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | |
| | Study product temperature excursion | | | | | | | | |
| | Other | | | | | | | | |
| Blinding policy/procedure | Any type | | | | | | | | |
| | Treatment unblinded | | | | | | | | |
| | Other | | | | | | | | |
| N=Number of enrolle | d subjects. | • | • | | | | | | • |

### 12.2.2 Displays of Adverse Events

# **Solicited Adverse Event Grading Scale**

Table 3: Local (Injection Site) Reactogenicity Grading

| Local (Injection Site)<br>Reaction | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
|---|---|---|---|
| Pain – experienced<br>without touching the<br>injection site<br>(spontaneous<br>discomfort) | Subject is aware of pain, but it does not interfere with daily activity, <b>and</b> no pain medication is taken | There is interference with daily activity <b>or</b> it requires repeated use of a non-narcotic pain reliever for >24 hours | Pain prevents daily<br>activity or requires any<br>use of a narcotic pain<br>reliever |
| Tenderness – hurts<br>only when injection<br>site is touched or the<br>arm is moved | hurts The area immediately The area cection surrounding the surrounding the injection site hurts only injection | | The area immediately surrounding the injection site hurts when touched or with arm motion, and it prevents daily activity |
| Pruritus (Itching) | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Ecchymosis (Bruising)* | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Erythema (Redness)* | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Induration (Hardness)/Swelling* | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |

<sup>\*</sup> Will also be measured in mm but size will not be used as halting criteria.

**Table 4:** Local (Injection Site) Reactogenicity Measurements

| Local (Injection Site) Reaction | Small | Medium | Large |
|---------------------------------|--------|---------------|--------|
| Ecchymosis (Bruising)* | <20 mm | 20 mm – 50 mm | >50 mm |
| Erythema (Redness)* | <20 mm | 20 mm – 50 mm | >50 mm |
| Induration (Hardness)/Swelling* | <20 mm | 20 mm – 50 mm | >50 mm |

<sup>\*</sup> Will not be used as halting criteria.

Table 5: Subjective Systemic Reactogenicity Grading

| Systemic (Subjective) | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
|---|---|---|---|
| Feverishness<br>(Chills/Shivering/Sweating) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Fatigue (Tiredness) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Malaise (General Unwell<br>Feeling) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Myalgia (Body<br>Aches/Muscular Pain)* | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |

| Systemic (Subjective) | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
|---|---|---|---|
| Arthralgia (Joint Pain)* | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Headache | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Nausea | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |

<sup>\*</sup> Not at injection site.

**Table 6: Quantitative Systemic Reactogenicity Grading** 

| Systemic (Quantitative) | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
|---|---|---|---|
| Fever* - oral† | 38.0°C – 38.4°C | 38.5°C – 38.9°C | >38.9°C |
| | 100.4°F – 101.1°F | 101.2°F – 102.0°F | >102.0°F |

Note: Oral temperature assessed on Day 1 prior to the first study vaccination will be considered as baseline.

**Table 7:** Additional Adverse Event Severity Grading

| Physiologic Parameter | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
|---|---|---|---|
| Bradycardia - beats per minute | 45 – 49 | 40 - 44 | <40 |
| Tachycardia - beats per minute | 116 – 130 | 131 – 155 | >155 |
| Hypotension (systolic) mm Hg | 80 - 84 | 75 – 79 | <75 |
| Hypotension (diastolic) mm Hg | 50 – 54 | 45 – 49 | <45 |
| Hypertension (systolic) mm Hg | 151 – 155 | 156 – 160 | >160 |
| Hypertension (diastolic) mm Hg | 96 – 100 | 101 – 105 | >105 |

<sup>\*</sup> A fever can be considered not related to the study product if an alternative etiology can be documented.

<sup>†</sup> Subjects must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.

## 14.1 Description of Study Subjects

## 14.1.1 Disposition of Subjects

Table 8: Subject Disposition by Treatment Group – All Enrolled Subjects

| Subject<br>Disposition | Study Arm 1 A/H3N2v,<br>D1 (N=X) | | • | /H7N9 + AS03,<br>(N=X) | Study Arm 3 A/H7N9 + PBS,<br>D1, 29 (N=X) | |
|---|---|---|---|---|---|---|
| | n | % | n | % | n | % |
| Screened | X | | X | | X | |
| Enrolled/Randomized | X | 100 | X | 100 | X | 100 |
| Received One Treatment | Х | xx | Х | XX | X | XX |
| Received All Scheduled Treatments <sup>a</sup> | X | xx | X | XX | X | XX |
| Completed Day 2 Omics Blood Draw | х | xx | Х | XX | X | xx |
| Completed Day 4 Omics Blood Draw | X | xx | X | XX | X | XX |
| Completed Day 8 Omics Blood Draw | х | xx | n/a | n/a | n/a | n/a |
| Completed Day 29 Omics Blood Draw | n/a | n/a | X | XX | X | XX |
| Completed Day 30 Omics Blood Draw | n/a | n/a | X | XX | X | XX |
| Completed Day 32 Omics Blood Draw | n/a | n/a | Х | XX | X | XX |
| Completed Day 36 Omics Blood Draw | n/a | n/a | X | XX | X | xx |
| Completed Follow-up (Study Day 29) <sup>a</sup> | | | n/a | n/a | n/a | n/a |
| Completed Follow-up (Study Day 366) <sup>a</sup> | n/a | n/a | X | XX | X | xx |
| Completed Per Protocol <sup>b</sup> | X | xx | X | XX | X | XX |

N=number of enrolled subjects

<sup>&</sup>lt;sup>a</sup> Refer to Listing of Early Terminations or Discontinued Subjects for reasons subjects discontinued or terminated early.

<sup>&</sup>lt;sup>b</sup> Refer to Listing of Analysis Populations Exclusions for reasons subjects are excluded from the Analysis populations.

Table 9: Analysis Populations by Treatment Group and Time Point – All Enrolled Subjects

| Analysis<br>Populations | Time Point Reason Subjects Excluded | | Study Arm 1<br>(A/H3N2v, D1)<br>(N=X) | | Study Arm 1<br>(A/H3N2v, D1)<br>(N=X) | | Group 3 3.75 µg A/H7N9 + PBS (D1, 29) (N=X) | |
|---|---|---|---|---|---|---|---|---|
| | | | n | % | n | % | % | n |
| Safety Analysis<br>Population | Any Time Point | Any Reason | х | XX | Х | xx | х | XX |
| | | [Reason 1, for example: Did not meet eligibility criteria] | | | | | | |
| | | [Reason 2] | | | | | | |
| | | [Reason 3] | | | | | | |
| | | [Reason 4] | | | | | | |
| ITT Analysis<br>Population | Any Time Point | Any Reason | | | | | | |
| | | [Reason 1] | | | | | | |
| | | [Reason 2] | | | | | | |
| PP Analysis<br>Population | Any Time Point | Any Reason | | | | | | |
| | | [Reason 1] | | | | | | |
| | | [Reason 2] | | | | | | |
| | Day 29 (Post-<br>Vaccination 1) | Any Reason | | | | | | |
| | | [Reason 1, for example: Did not meet eligibility criteria] | | | | | | |
| | | [Reason 2] | | | | | | |
| | | [Reason 3] | | | | | | |

**Table 10:** Ineligibility Summary of Screen Failures

| Inclusion/Exclusion Category | Inclusion/Exclusion Criterion | n <sup>a</sup> | <b>⁰∕₀</b> b |
|---|---|---|---|
| Inclusion and Exclusion | Number of subjects failing any eligibility criterion | X | XX |
| Inclusion | Any inclusion criterion | X | XX |
| | [inclusion criterion 1] | X | XX |
| | [inclusion criterion 2] | X | XX |
| | [inclusion criterion 3] | X | XX |
| Exclusion | Any exclusion criterion | X | XX |
| | [exclusion criterion 1] | X | XX |
| | [exclusion criterion 2] | X | XX |
| | [exclusion criterion 3] | X | XX |
| Eligible but not enrolled | | X | XX |

<sup>&</sup>lt;sup>a</sup> More than one criterion may be marked per subject.

<sup>&</sup>lt;sup>b</sup>Denominator for percentages is the total number of screen failures.

# 14.1.2 Demographic Data by Study Group

Table 11: Summary of Categorical Demographic and Baseline Characteristics by Treatment Group - All Enrolled Subjects

| Variable | Characteristic | Study Arm 1<br>A/H3N2v, D1 (N=X) | | Study Arm 2<br>A/H7N9 + AS03,<br>D1, 29 (N=X) | | Study Arm 3<br>A/H7N9 +<br>PBS, D1, 29<br>(N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % |
| Sex | Male | x | xx | x | XX | х | XX | х | xx |
| | Female | | | | | | | | |
| Ethnicity | Not Hispanic or Latino | х | xx | х | xx | х | xx | Х | XX |
| | Hispanic or Latino | | | | | | | | |
| | Not Reported | | | | | | | | |
| | Unknown | | | | | | | | |
| Race | American Indian or Alaska Native | х | xx | x | xx | х | XX | х | xx |
| | Asian | | | | | | | | |
| | Native Hawaiian or Other Pacific<br>Islander | | | | | | | | |
| | Black or African American | | | | | | | | |
| | White | | | | | | | | |
| | Multi-Racial | | | | | | | | |
| | Unknown | | | | | | | | |
| N=Number of 6 | enrolled subjects. | • | • | • | • | • | | • | • |

Table 12: Summary of Continuous Demographic and Baseline Characteristics by Treatment Group - All Enrolled Subjects

| Variable | Statistic | Study Arm 1<br>A/H3N2v, D1<br>(N=X) | Study Arm 2 A/H7N9<br>+ AS03, D1, 29 (N=X) | Study Arm 3<br>A/H7N9 + PBS,<br>D1, 29 (N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|
| Age (units) | Mean | x x | x.x | x.x | x x |
| | Standard Deviation | хх | X.X | x.x | хх |
| | Median | X | X | X | X |
| | Minimum | X | X | Х | X |
| | Maximum | X | X | X | X |
| BMI | Mean | x x | x.x | x.x | хх |
| | Standard Deviation | x x | X.X | x.x | хх |
| | Median | X | X | Х | х |
| | Minimum | X | X | Х | X |
| | Maximum | x | X | Х | Х |
| N=Number of enroll | ed subjects. | | • | | |

#### 14.1.3 Prior and Concurrent Medical Conditions

Table 13: Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group

| MedDRA System Organ Class | | Study Arm 1<br>A/H3N2v, D1 (N=X) | | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) | | Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|---|---|
| | n | % | n | % | n | % | n | % |
| Any SOC | x | xx | X | XX | X | xx | х | xx |
| [SOC 1] | | | | | | | | |
| [SOC 2] | | | | | | | | |

Note: N=Number of subjects in the Safety Population

n = Number of subjects reporting medical history within the specified SOC. A subject is only counted once per SOC.

#### 14.2 Immunogenicity Data

#### 14.2.1 Serum Antibody Data

Table 14: Summaries of Hemagglutination Inhibition Antibody Titer by Study Day and Treatment Group in the Intent-to-Treat Population

| Time Point | Statistic | Study Arm 1<br>A/H3N2v, D1 (N=X) | Study Arm 2<br>A/H7N9 + AS03, D1,<br>29 (N=X) | Study Arm 3 A/H7N9<br>+ PBS, D1, 29 (N=X) |
|---|---|---|---|---|
| Day 1 (Pre-Vaccination 1) | n | X | X | X |
| | GMT (95% CI) | x x (x.x,x x) | x.x (x x,x.x) | x x (x x,x.x) |
| Day 29 (Post-Vaccination 1) | n | х | X | X |
| | GMT (95% CI) | x x (x.x,x x) | x.x (x x,x.x) | x x (x x,x.x) |
| | Seroconversion n/N (%) [95% CI] | xx/xx (xx%) [xx, xx] | xx/xx (xx%) [xx, xx] | xx/xx (xx%) [xx, xx] |
| Day 29 (Post-Vaccination 2) | n | n/a | х | Х |
| | GMT (95% CI) | n/a | x.x (x x,x.x) | x x (x x,x.x) |
| | Seroconversion n/N (%) [95%<br>CI] | n/a | xx/xx (xx%) [xx, xx] | xx/xx (xx%) [xx, xx] |

N = Number of subjects in the Intent-to-Treat Population

Seroconversion is defined as having a pre -vaccination titer  $\le 1:10$  and a post - vaccination titer  $\ge 1:40$  or a pre - vaccination titer  $\ge 1:10$  and a minimum four -fold rise in post-vaccination antibody titer

- Table 15: Summaries of Hemagglutination Inhibition Antibody Titer by Study Day and Treatment Group in the Per-Protocol Population
- Table 16: Summaries of Neutralizing Antibody by Study Day and Treatment Group in the Intentto-Treat Population
- Table 17: Summaries of Neutralizing Antibody by Study Day and Treatment Group in the Per-Protocol Population

n = Number of subjects with available results

GMT = Geometric mean titer

Table 18: t-Test Results for Comparing Day 29 Post-Last Vaccination Hemagglutination Inhibition Antibody Titer between Treatment Groups in the Intent-to-Treat Population

| Statistic | Study Arm 2<br>A/H7N9 + AS03, D1, 29 (N=X)<br>vs. Study Arm 3 A/H7N9 +<br>PBS, D1, 29 (N=X) | Study Arm 2<br>A/H7N9 + AS03, D1, 29 (N=X)<br>vs. Study Arm 1<br>A/H3N2v, D1 (N=X) | Study Arm 3 A/H7N9 + PBS,<br>D1, 29 (N=X) vs.<br>Study Arm 1<br>A/H3N2v, D1 (N=X) |
|---|---|---|---|
| n | xx | XX | XX |
| GMT Ratio (95% CI) | x xx (x xx,x xx) | x xx (x xx,x xx) | x.xx (x.xx,x.xx) |
| t-statistic | x xxx | x.xxx | x xxx |
| P-value | x xxx | x.xxx | x xxx |

N = Number of subjects in the Intent-to-Treat Population

- Table 19: t-Test Results for Comparing Day 29 Post-Last Vaccination Hemagglutination Inhibition
  Antibody Titer Between Treatment Groups in the Per-Protocol Population
- Table 20: t-Test Results for Comparing Day 29 Post-Last Vaccination Neutralizing Antibody Titer Between Treatment Groups in the Intent-to-Treat Population
- Table 21: t-Test Results for Comparing Day 29 Post-Last Vaccination Neutralizing Antibody Titer Between Treatment Groups in the Per-Protocol Population

n = Number of subjects with available results

P-value = two-sided Welch's or standard t-test P-value

Table 22: Fisher's Exact Test Results for Comparing Day 29 Post-Last Vaccination Seroconversion based on Hemagglutination Inhibition Antibody Titer Between Treatment Groups in the Intent-to-Treat Population

| | Study Arm 2<br>A/H7N9 + AS03, D1, 29 (N=X) vs. Study<br>Arm 3 A/H7N9 + PBS, D1, 29 (N=X) | Study Arm 2<br>A/H7N9 + AS03, D1, 29 (N=X) vs. Study<br>Arm 1<br>A/H3N2v, D1 (N=X) | Study Arm 3 A/H7N9 + PBS, D1, 29 (N=X) vs. Study Arm 1 A/H3N2v, D1 (N=X) |
|---|---|---|---|
| n | xx | XX | xx |
| Seroconversion n/N (%) [95% CI] | xx/xx (xx%) [xx, xx] | xx/xx (xx%) [xx, xx] | xx/xx (xx%) [xx, xx] |
| Exact Odds Ratio(95% CI) | x.xxx | x xxx | x.xxx |
| p-value | x.xxx | x xxx | x.xxx |

N = Number of subjects in the Intent-to-Treat Population

P-value = two-sided Fisher's Exact test P-vale.

- Table 23: Fisher's Exact Test Results for Comparing Day 29 Post-Last Vaccination Seroconversion based on Hemagglutination Inhibition Antibody Titer Between Treatment Groups in the Per-Protocol Population
- Table 24: Fisher's Exact Test Results for Comparing Day 29 Post-Last Vaccination Seroconversion based on Neutralizing Antibody between Treatment Groups in the Intent-to-Treat Population
- Table 25: Fisher's Exact Test Results for Comparing Day 29 Post-Last Vaccination Seroconversion based on Neutralizing Antibody between Treatment Groups in the Per-Protocol Population

n = Number of subjects with available results

## 14.2.2 Plasma Cytokine/Chemokine Data

Table 26: Fractalkine Concentration by Study Visit Day and Treatment Group in the Intent-to-Treat Population

| Time Point | Statistic | Study Arm 1<br>A/H3N2v, D1<br>(N=X) | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) | Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) |
|---|---|---|---|---|
| Day 1 (Pre-Vaccination 1) | n | X | x | X |
| | Min | x xx | x xx | x xx |
| | Q1 | X X | x.x | хх |
| | Median (95% CI) | x x (x x - x.x) | x.x (x x - x.x) | x x (x x - x x) |
| | Q3 | X X | x.x | хх |
| | Max | x xx | x xx | x xx |
| Day 2 (Post-Vaccination 1) | n | X | X | X |
| | Min | x xx | x xx | x xx |
| | Q1 | X X | X.X | хх |
| | Median (95% CI) | x x (x x - x.x) | x.x (x x - x.x) | x x (x x - x x) |
| | Q3 | X X | x.x | хх |
| | Max | x xx | x xx | x xx |
| Day 4 (Post-Vaccination 1) | n | X | X | X |
| | Min | x xx | x xx | x xx |
| | Q1 | X X | x.x | хх |
| | Median (95% CI) | x x (x x - x.x) | x.x (x x - x.x) | x x (x x - x x) |
| | Q3 | X X | x.x | хх |
| | Max | x xx | x xx | x xx |
| Day 8 (Post-Vaccination 1) | n | X | n/a | n/a |
| | Min | x xx | n/a | n/a |
| | Q1 | X X | n/a | n/a |
| | Median (95% CI) | x x (x x - x.x) | n/a | n/a |
| | Q3 | X X | n/a | n/a |

| Time Point | Statistic | Study Arm 1<br>A/H3N2v, D1<br>(N=X) | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) | Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) |
|---|---|---|---|---|
| | Max | x xx | n/a | n/a |
| Day 29 (Post-Vaccination 1) | n | n/a | x | X |
| | Min | n/a | x xx | X XX |
| | Q1 | n/a | X.X | хх |
| | Median (95% CI) | n/a | x.x (x x - x.x) | x x (x x - x x) |
| | Q3 | n/a | x.x | хх |
| | Max | n/a | x xx | x xx |
| Day 2 (Post-Vaccination 2) | n | n/a | x | X |
| | Min | n/a | x xx | x xx |
| | Q1 | n/a | x.x | X X |
| | Median (95% CI) | n/a | x.x (x x - x.x) | x x (x x - x x) |
| | Q3 | n/a | x.x | X X |
| | Max | n/a | x xx | X XX |
| Day 4 (Post-Vaccination 2) | n | n/a | x | X |
| | Min | n/a | x xx | x xx |
| | Q1 | n/a | x.x | хх |
| | Median (95% CI) | n/a | x.x (x x - x.x) | x x (x x - x x) |
| | Q3 | n/a | x.x | хх |
| | Max | n/a | x xx | x xx |
| Day 8 (Post-Vaccination 2) | n | n/a | x | X |
| | Min | n/a | x xx | X XX |
| | Q1 | n/a | X.X | хх |
| | Median (95% CI) | n/a | x.x (x x - x.x) | x x (x x - x x) |
| | Q3 | n/a | X.X | хх |
| | Max | n/a | x xx | x xx |

| Time Point | Statistic | Study Arm 1<br>A/H3N2v, D1 | Study Arm 2<br>A/H7N9 + AS03, D1, 29 | Study Arm 3<br>A/H7N9 + PBS, D1, 29 |
|---|---|---|---|---|
| | | (N=X) | (N=X) | (N=X) |

N= Number of subjects in the Intent-to-Treat analysis population n= Number of subjects with valid results

Min=Minimum

Q1= First quartile

Q3=Third quartile

Max=Maximum

The 95% CI of the median is based on the bootstrap method.

| <b>Table 27:</b> | Fractalkine Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population |
|---|---|
| Table 28: | GM-CSF Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population |
| Table 29: | GM-CSF Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population |
| Table 30: | Interferon-gamma Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population |
| Table 31: | Interferon-gamma Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population |
| <b>Table 32:</b> | Interleukin 1 beta Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population |
| Table 33: | Interleukin 1 beta Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population |
| Table 34: | Interleukin 2 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population |
| <b>Table 35:</b> | Interleukin 2 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population |
| Table 36: | Interleukin 4 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population |
| <b>Table 37:</b> | Interleukin 4 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population |
| Table 38: | Interleukin 5 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population |
| Table 39: | Interleukin 5 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population |
| Table 40: | Interleukin 6 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population |
| Table 41: | Interleukin 6 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population |
| Table 42: | Interleukin 7 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population |

Table 43: Interleukin 7 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population Table 44: Interleukin 8 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 45:** Interleukin 8 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population Interleukin 10 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population Table 46: **Table 47:** Interleukin 10 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population Table 48: Interleukin-12, p70 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population Table 49: Interleukin-12, p70 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population Table 50: Interleukin 13 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 51:** Interleukin 13 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 52:** IL-17A Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 53:** IL-17A Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 54:** Interleukin 21 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 55:** Interleukin 21 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 56:** Interleukin 23 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 57:** Interleukin 23 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 58:** Interferon-inducible T Cell Alpha Chemoattractant Concentration by Study Visit Day and Treatment Group in the Intent-To-**Treat Population Table 59:** Interferon-inducible T Cell Alpha Chemoattractant Concentration by Study Visit Day and Treatment Group in the Per-Protocol **Population** Table 60: Macrophage Inflammatory Protein 1 Alpha Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat **Population** Table 61: Macrophage Inflammatory Protein 1 Alpha Concentration by Study Visit Day and Treatment Group in the Per-Protocol **Population** 

Macrophage Inflammatory Protein-1 Beta Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Table 62: **Population** Table 63: Macrophage Inflammatory Protein-1 Beta Concentration by Study Visit Day and Treatment Group in the Per-Protocol **Population** Macrophage Inflammatory Protein-3 Alpha Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Table 64: **Population Table 65:** Macrophage Inflammatory Protein-3 Alpha Concentration by Study Visit Day and Treatment Group in the Per-Protocol **Population** Tumor Necrosis Factor Alpha Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population Table 66: Tumor Necrosis Factor Alpha Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population Table 67: Table 68: Interferon Gamma-Induced Protein 10 Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat **Population** Table 69: Interferon Gamma-Induced Protein 10 Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 70:** Interferon-Alpha Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 71:** Interferon-Alpha Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population Interferon-Beta Concentration by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 72:** Interferon-Beta Concentration by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 73:** 

Table 74: Fractalkine Fold Change by Study Visit Day and Study Group in the Intent-To-Treat Population

| Time Point | Statistic | Study Arm 1<br>A/H3N2v, D1<br>(N=X) | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) | Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) |
|---|---|---|---|---|
| Day 2 (Post-Vaccination 1) | n | X | x | X |
| | Min | x xx | x xx | X XX |
| | Q1 | x x | x.x | X X |
| | Median (95% CI) | x x (x x - x.x) | x.x (x x - x.x) | x x (x x - x x) |
| | Q3 | x x | x.x | хх |
| | Max | x xx | x xx | x xx |
| Day 4 (Post-Vaccination 1) | n | X | x | X |
| | Min | x xx | x xx | x xx |
| | Q1 | x x | x.x | x x |
| | Median (95% CI) | x x (x x - x.x) | x.x (x x - x.x) | x x (x x - x x) |
| | Q3 | x x | x.x | хх |
| | Max | x xx | x xx | x xx |
| Day 8 (Post-Vaccination 1) | n | X | n/a | n/a |
| | Min | x xx | n/a | n/a |
| | Q1 | x x | n/a | n/a |
| | Median (95% CI) | x x (x x - x.x) | n/a | n/a |
| | Q3 | x x | n/a | n/a |
| | Max | x xx | n/a | n/a |
| Day 29 (Post-Vaccination 1) | n | n/a | x | X |
| | Min | n/a | x xx | x xx |
| | Q1 | n/a | X.X | X X |
| | Median (95% CI) | n/a | x.x (x x - x.x) | x x (x x - x x) |
| | Q3 | n/a | X.X | X X |
| | Max | n/a | x xx | x xx |

| Time Point | Statistic | Study Arm 1<br>A/H3N2v, D1<br>(N=X) | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) | Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) |
|---|---|---|---|---|
| Day 2 (Post-Vaccination 2) | n | n/a | x | Х |
| | Min | n/a | x xx | x xx |
| | Q1 | n/a | X.X | хх |
| | Median (95% CI) | n/a | x.x (x x - x.x) | x x (x x - x x) |
| | Q3 | n/a | X.X | хх |
| | Max | n/a | x xx | x xx |
| Day 4 (Post-Vaccination 2) | n | n/a | x | х |
| | Min | n/a | x xx | x xx |
| | Q1 | n/a | x.x | хх |
| | Median (95% CI) | n/a | x.x (x x - x.x) | x x (x x - x x) |
| | Q3 | n/a | x.x | хх |
| | Max | n/a | x xx | X XX |
| Day 8 (Post-Vaccination 2) | n | n/a | x | Х |
| | Min | n/a | x xx | X XX |
| | Q1 | n/a | x.x | хх |
| | Median (95% CI) | n/a | x.x (x x - x.x) | x x (x x - x x) |
| | Q3 | n/a | x.x | хх |
| | Max | n/a | x xx | X XX |

N= Number of subjects in the Intent-to-Treat population n= Number of subjects with valid results

Min=Minimum

Q1= First quartile Q3=Third quartile

Max=Maximum

The 95% CI of the median is based on the bootstrap method.

#### Tables with similar format:

**Table 75:** Fractalkine Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 76:** GM-CSF Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 77:** GM-CSF Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 78:** Interferon-gamma Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 79:** Interferon-gamma Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population Table 80: Interleukin 1 beta Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 81:** Interleukin 1 beta Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 82:** Interleukin 2 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 83:** Interleukin 2 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 84:** Interleukin 4 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 85:** Interleukin 4 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 86:** Interleukin 5 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 87:** Interleukin 5 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 88:** Interleukin 6 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 89:** Interleukin 6 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population Table 90: Interleukin 7 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population Table 91: Interleukin 7 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population Interleukin 8 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population Table 92: Table 93: Interleukin 8 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population Table 94: Interleukin 10 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 95:** Interleukin 10 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population Table 96: Interleukin-12, p70 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 97:** Interleukin-12, p70 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population

Table 98: Interleukin 13 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population Table 99: Interleukin 13 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 100:** IL-17A Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 101:** IL-17A Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 102:** Interleukin 21 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 103:** Interleukin 21 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 104:** Interleukin 23 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population Interleukin 23 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 105: Table 106:** Interferon-inducible T Cell Alpha Chemoattractant Fold Change by Study Visit Day and Treatment Group in the Intent-To-**Treat Population Table 107:** Interferon-inducible T Cell Alpha Chemoattractant Fold Change by Study Visit Day and Treatment Group in the Per-Protocol **Population Table 108:** Macrophage Inflammatory Protein 1 Alpha Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat **Population** Macrophage Inflammatory Protein 1 Alpha Fold Change by Study Visit Day and Treatment Group in the Per-Protocol **Table 109: Population** Macrophage Inflammatory Protein-1 Beta Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat **Table 110: Population Table 111:** Macrophage Inflammatory Protein-1 Beta Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population Macrophage Inflammatory Protein-3 Alpha Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat **Table 112: Population Table 113:** Macrophage Inflammatory Protein-3 Alpha Fold Change by Study Visit Day and Treatment Group in the Per-Protocol **Population** Tumor Necrosis Factor Alpha Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 114:** Tumor Necrosis Factor Alpha Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population **Table 115:** Interferon Gamma-Induced Protein 10 Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population **Table 116:**
- Table 117: Interferon Gamma-Induced Protein 10 Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population
- Table 118: Interferon-Alpha Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population
- Table 119: Interferon-Alpha Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population
- Table 120: Interferon-Beta Fold Change by Study Visit Day and Treatment Group in the Intent-To-Treat Population
- Table 121: Interferon-Beta Fold Change by Study Visit Day and Treatment Group in the Per-Protocol Population

Table 122: Wilcoxon Signed-Rank Test Results for Comparing Cytokine/Chemokine Concentrations between Pre- and Post-Vaccination Time Points in the Intent-To-Treat Population

| | | Study Arm 1<br>A/H3N2v, D1<br>(N=X) | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) | Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) |
|---|---|---|---|---|
| Cytokine | Comparison | Wilcoxon Statistic<br>(P-value) | Wilcoxon Statistic<br>(P-value) | Wilcoxon Statistic<br>(P-value) |
| Fractalkine | Day 2 (Post -Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x xxx) | x xxx (x xxx) | x.xxx (x xxx) |
| Fractalkine | Day 4 (Post-Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x.xxx) | x xxx (x xxx) | x.xxx (x xxx) |
| Fractalkine | Day 8 (Post-Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x.xxx) | n/a | n/a |
| Fractalkine | Day 29 (Post-Vaccination 1) vs. Pre-Vaccination 1 | n/a | x xxx (x xxx) | x.xxx (x xxx) |
| Fractalkine | Day 2 (Post-Vaccination 2) vs. Pre-Vaccination 2 | n/a | x xxx (x xxx) | x.xxx (x xxx) |
| Fractalkine | Day 4 (Post-Vaccination 2) vs. Pre-Vaccination 2 | n/a | x xxx (x xxx) | x.xxx (x xxx) |
| Fractalkine | Day 8 (Post-Vaccination 2) vs. Pre-Vaccination 2 | n/a | x xxx (x xxx) | x.xxx (x xxx) |
| GM-CSF | Day 2 (Post -Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x xxx) | x xxx (x xxx) | x.xxx (x xxx) |
| GM-CSF | Day 4 (Post-Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x.xxx) | x xxx (x xxx) | x.xxx (x xxx) |
| GM-CSF | Day 8 (Post-Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x.xxx) | n/a | n/a |
| GM-CSF | Day 29 (Post-Vaccination 1) vs. Pre-Vaccination 1 | n/a | x xxx (x xxx) | x.xxx (x xxx) |
| GM-CSF | Day 2 (Post-Vaccination 2) vs. Pre-Vaccination 2 | n/a | x xxx (x xxx) | x.xxx (x xxx) |
| GM-CSF | Day 4 (Post-Vaccination 2) vs. Pre-Vaccination 2 | n/a | x xxx (x xxx) | x.xxx (x xxx) |
| GM-CSF | Day 8 (Post-Vaccination 2) vs. Pre-Vaccination 2 | n/a | x xxx (x xxx) | x.xxx (x xxx) |
| Interferon-gamma | Day 2 (Post -Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x xxx) | x xxx (x xxx) | x.xxx (x xxx) |
| Interferon-gamma | Day 4 (Post-Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x.xxx) | x xxx (x xxx) | x.xxx (x xxx) |
| Interferon-gamma | Day 8 (Post-Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x.xxx) | n/a | n/a |
| Interferon-gamma | Day 29 (Post-Vaccination 1) vs. Pre-Vaccination 1 | n/a | x xxx (x xxx) | x.xxx (x xxx) |
| Interferon-gamma | Day 2 (Post-Vaccination 2) vs. Pre-Vaccination 2 | n/a | x xxx (x xxx) | x.xxx (x xxx) |
| Interferon-gamma | Day 4 (Post-Vaccination 2) vs. Pre-Vaccination 2 | n/a | x xxx (x xxx) | x.xxx (x xxx) |
| Interferon-gamma | Day 8 (Post-Vaccination 2) vs. Pre-Vaccination 2 | n/a | x xxx (x xxx) | x.xxx (x xxx) |
| Colored in blue= p-v | alue < 0.05 | | · · | |

Continue for the remaining cytokine/chemokines IL-1b, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12p70, IL-13, IL-17A, IL-21, IL-23, ITAC, MIP 1a, MIP1b, MIP3a, TNF-alpha, IP-10, IFNa, IFNb Table with similar format:

Table 123: Wilcoxon Signed-Rank Test Results for Comparing Cytokine/Chemokine Concentrations between Pre- and Post-Vaccination Time Points in the Per-Protocol Population

Table 124: Wilcoxon Rank Sum Test Results for Comparing Fold Changes between Study Groups in the Intent-To-Treat Population

| | | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) vs.<br>Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) vs.<br>Study Arm 1<br>A/H3N2v, D1<br>(N=X) | Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) vs.<br>Study Arm 1<br>A/H3N2v, D1<br>(N=X) |
|---|---|---|---|---|
| Cytokine | Comparison | Wilcoxon Statistic<br>(p-value) | Wilcoxon Statistic<br>(p-value) | Wilcoxon Statistic<br>(p-value) |
| Fractalkine | Day 2 (Post -Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x xxx) | x xxx (x xxx) | x.xxx (x xxx) |
| Fractalkine | Day 4 (Post-Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x xxx) | x xxx (x xxx) | x.xxx (x xxx) |
| Fractalkine | Day 29 (Post-Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x xxx) | n/a | n/a |
| Fractalkine | Day 2 (Post-Vaccination 2) vs. Pre-Vaccination 2 | x xxx (x xxx) | n/a | n/a |
| Fractalkine | Day 4 (Post-Vaccination 2) vs. Pre-Vaccination 2 | x xxx (x xxx) | n/a | n/a |
| Fractalkine | Day 8 (Post-Vaccination 2) vs. Pre-Vaccination 2 | x xxx (x xxx) | n/a | n/a |
| GM-CSF | Day 2 (Post -Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x xxx) | x xxx (x xxx) | x.xxx (x xxx) |
| GM-CSF | Day 4 (Post-Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x xxx) | x xxx (x xxx) | x.xxx (x xxx) |
| GM-CSF | Day 29 (Post-Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x xxx) | n/a | n/a |
| GM-CSF | Day 2 (Post-Vaccination 2) vs. Pre-Vaccination 2 | x xxx (x xxx) | n/a | n/a |
| GM-CSF | Day 4 (Post-Vaccination 2) vs. Pre-Vaccination 2 | x xxx (x xxx) | n/a | n/a |
| GM-CSF | Day 8 (Post-Vaccination 2) vs. Pre-Vaccination 2 | x xxx (x xxx) | n/a | n/a |
| Interferon-gamma | Day 2 (Post -Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x xxx) | x xxx (x xxx) | x.xxx (x xxx) |
| Interferon-gamma | Day 4 (Post-Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x xxx) | x xxx (x xxx) | x.xxx (x xxx) |
| Interferon-gamma | Day 29 (Post-Vaccination 1) vs. Pre-Vaccination 1 | x xxx (x xxx) | n/a | n/a |
| Interferon-gamma | Day 2 (Post-Vaccination 2) vs. Pre-Vaccination 2 | x xxx (x xxx) | n/a | n/a |
| Interferon-gamma | Day 4 (Post-Vaccination 2) vs. Pre-Vaccination 2 | x xxx (x xxx) | n/a | n/a |
| Interferon-gamma | Day 8 (Post-Vaccination 2) vs. Pre-Vaccination 2 | x xxx (x xxx) | n/a | n/a |
| Colored in blue= p-va | alue < 0.05 | | | |

Continue for the remaining cytokine/chemokines IL-1b, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12p70, IL-13, IL-17A, IL-21, IL-23, ITAC, MIP 1a, MIP1b, MIP3a, TNF-alpha, IP-10, IFNa, IFNb

Table with similar format:

Table 125: Wilcoxon Rank Sum Test Results for Comparing Fold Changes between Study Groups in the Per-Protocol Population

### 14.3 Transcriptomics Data

Table 126: Genes Differentially Expressed Compared to Pre-Vaccination by Treatment Group, Cell Type, and Post-Vaccination Day

| | | Study Arm 1<br>A/H3N2v, D1<br>(N=X) | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) | Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) |
|---|---|---|---|---|
| Time Point | Cell Type | DE Genes [#] | DE Genes [#] | DE Genes [#] |
| Day 2 (Post Vaccination 1 vs. Pre-Vaccination 1) | Monocytes | xxx | XXX | XXX |
| | Dendritic cells | xxx | XXX | XXX |
| | Neutrophils | xxx | xxx | XXX |
| | NK-cells | XXX | XXX | XXX |
| | T-cells | XXX | XXX | XXX |
| | B-cells | XXX | XXX | XXX |
| Day 4 (Post Vaccination 1 vs. Pre-Vaccination 1) | Monocytes | XXX | XXX | XXX |
| | Dendritic cells | xxx | xxx | XXX |
| | Neutrophils | XXX | XXX | XXX |
| | NK-cells | XXX | xxx | XXX |
| | T-cells | xxx | xxx | XXX |
| | B-cells | XXX | xxx | XXX |
| Day 8 (Post Vaccination 1 vs. Pre-Vaccination 1) | Monocytes | xxx | n/a | n/a |
| | Dendritic cells | xxx | n/a | n/a |
| | Neutrophils | xxx | n/a | n/a |
| | NK-cells | XXX | n/a | n/a |
| | T-cells | xxx | n/a | n/a |
| | B-cells | xxx | n/a | n/a |
| Day 29 (Post Vaccination 1 vs. Pre-Vaccination 1) | Monocytes | n/a | xxx | XXX |
| | Dendritic cells | n/a | xxx | XXX |
| | Neutrophils | n/a | xxx | XXX |
| | NK-cells | n/a | xxx | XXX |

| | | Study Arm 1<br>A/H3N2v, D1<br>(N=X) | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) | Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) |
|---|---|---|---|---|
| | T-cells | n/a | XXX | XXX |
| | B-cells | n/a | xxx | XXX |
| Day 2 (Post Vaccination 2 vs. Pre-Vaccination 2) | Monocytes | n/a | xxx | XXX |
| | Dendritic cells | n/a | xxx | XXX |
| | Neutrophils | n/a | XXX | XXX |
| | NK-cells | n/a | XXX | XXX |
| | T-cells | n/a | XXX | XXX |
| | B-cells | n/a | xxx | XXX |
| Day 4 (Post Vaccination 2 vs. Pre-Vaccination 2) | Monocytes | n/a | XXX | XXX |
| | Dendritic cells | n/a | XXX | XXX |
| | Neutrophils | n/a | xxx | XXX |
| | NK-cells | n/a | xxx | XXX |
| | T-cells | n/a | xxx | XXX |
| | B-cells | n/a | xxx | XXX |
| Day 8 (Post Vaccination 2 vs. Pre-Vaccination 2) | Monocytes | n/a | XXX | XXX |
| | Dendritic cells | n/a | XXX | XXX |
| | Neutrophils | n/a | xxx | XXX |
| | NK-cells | n/a | xxx | XXX |
| | T-cells | n/a | xxx | XXX |
| | B-cells | n/a | XXX | XXX |

N=Number of subjects in the Omics analysis population DE Gene = differentially expressed gene

Genes Differentially Expressed Between Treatment Groups by Immune Cell Type, and Post-Vaccination Day **Table 127:** 

Table 127: Genes Differentially Expressed Between Treatment Groups by Immune Cell Type, and Post-Vaccination Day

| | | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) vs.<br>Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) vs.<br>Study Arm 1<br>A/H3N2v, D1<br>(N=X) | Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) vs.<br>Study Arm 1<br>A/H3N2v, D1<br>(N=X) |
|---|---|---|---|---|
| Time Point | Cell Type | DE Genes [#] | DE Genes [#] | DE Genes [#] |
| Day 2 (Post Vaccination 1 vs. Pre-Vaccination 1) | Monocytes | XXX | XXX | XXX |
| | Dendritic cells | xxx | xxx | XXX |
| | Neutrophils | xxx | xxx | xxx |
| | NK-cells | xxx | xxx | xxx |
| | T-cells | xxx | xxx | xxx |
| | B-cells | xxx | xxx | xxx |
| Day 4 (Post Vaccination 1 vs. Pre-Vaccination 1) | Monocytes | xxx | xxx | xxx |
| | Dendritic cells | xxx | xxx | xxx |
| | Neutrophils | xxx | xxx | xxx |
| | NK-cells | XXX | XXX | xxx |
| | T-cells | xxx | XXX | xxx |
| | B-cells | xxx | xxx | xxx |
| Day 29 (Post Vaccination 1 vs. Pre-Vaccination 1) | Monocytes | XXX | n/a | n/a |
| | Dendritic cells | xxx | n/a | n/a |
| | Neutrophils | xxx | n/a | n/a |
| | NK-cells | XXX | n/a | n/a |
| | T-cells | XXX | n/a | n/a |
| | B-cells | XXX | n/a | n/a |
| Day 2 (Post Vaccination 2 vs. Pre-Vaccination 2) | Monocytes | XXX | n/a | n/a |
| | Dendritic cells | xxx | n/a | n/a |

| | | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) vs.<br>Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) vs.<br>Study Arm 1<br>A/H3N2v, D1<br>(N=X) | Study Arm 3 A/H7N9 + PBS, D1, 29 (N=X) vs. Study Arm 1 A/H3N2v, D1 (N=X) |
|---|---|---|---|---|
| | Neutrophils | XXX | n/a | n/a |
| | NK-cells | xxx | n/a | n/a |
| | T-cells | xxx | n/a | n/a |
| | B-cells | XXX | n/a | n/a |
| Day 4 (Post Vaccination 2 vs. Pre-Vaccination 2) | Monocytes | XXX | n/a | n/a |
| | Dendritic cells | XXX | n/a | n/a |
| | Neutrophils | XXX | n/a | n/a |
| | NK-cells | XXX | n/a | n/a |
| | T-cells | XXX | n/a | n/a |
| | B-cells | XXX | n/a | n/a |
| Day 8 (Post Vaccination 2 vs. Pre-Vaccination 2) | Monocytes | XXX | n/a | n/a |
| | Dendritic cells | XXX | n/a | n/a |
| | Neutrophils | xxx | n/a | n/a |
| | NK-cells | XXX | n/a | n/a |
| | T-cells | XXX | n/a | n/a |
| | B-cells | xxx | n/a | n/a |

N=Number of subjects in the Omics analysis population DE Gene = differentially expressed gene

#### Table 128: Genes Differentially Expressed at Day 2 Compared to Pre-First Vaccination (RNA-Seq, Monocytes, Study Arm 1 A/H3N2v, D1)

Generate tables for each applicable post-vaccination day, treatment group, pairwise treatment group comparisons (Group 1 vs. 2, Group 1 vs. 3, Group 1 vs. 3, and Group 2 vs. 3), and cell type (monocytes, neutrophils, dendritic cells, NK cells B cell, and T cells). For Group 1 include tables for days 2, 4, and 8 post-first vaccination. For Groups 2 and 3 provide tables for post-vaccination days 2, 4, 29, 30, 32, and 36 post-first vaccination. For pairwise group comparisons that include Group 1, generate tables for days 2 and 4 post-first vaccination. Otherwise, prepare comparison results for days 2,4, 29, 30, 32, and 36 post-first vaccination.

| Ensembl<br>Gene ID | Ensembl<br>Gene Name | Ensembl<br>Gene Description | Gene<br>Type | Log <sub>2</sub> Fold Change<br>(Day 2 vs. Pre-First<br>Vaccination) | Average<br>Log <sub>2</sub><br>CPM* | Likelihood Ratio<br>Test Statistic | P-Value | FDR<br>Adjusted P-<br>value |
|---|---|---|---|---|---|---|---|---|
| ENSG00000<br>115415 | STAT1 | signal transducer and activator of transcription 1, 91kDa [Source:HGNC Symbol;Acc:11362] | protein coding | 1.94 | 2.034 | 5.324 | 0.000034 | 0.000613 |
| ENSG00000<br>125347 | IRF1 | interferon regulatory factor 1 [Source:HGNC<br>Symbol;Acc:6116] | protein<br>coding | 0.672 | 2.506 | 4.324 | 0.0343 | 0.00234 |
| ENSG00000<br>247275 | AL160008.1 | | lincRNA | 0.80 | 0.96 | 3.42 | 0.043 | 0.0483 |

<sup>\*:</sup> average gene expression levels across Day 2 and Pre-First Vaccination samples measured in average log2 CPM

### Table 129: Clusters of Co-Expressed Differential Genes (Monocytes, Days 2-29)

Generate tables for each fold change set (Day 2-29 post-first vaccination and Day 2-8 post-second vaccination) and cell type (monocytes, neutrophils, dendritic cells, NK cells B cell, and T cells)

| Cluster ID | Cluster Size | Ensembl<br>Gene ID | Ensembl Gene Name | Ensembl<br>Gene Description | Gene Type | KEGG Pathway |
|---|---|---|---|---|---|---|
| CCD229-001 | 3 | ENSG00000115415 | STAT1 | signal transducer and activator of transcription 1, 91kDa [Source:HGNC Symbol;Acc:11362] | protein coding | Jak-STAT signaling pathway |
| | | ENSG00000125347 | IRF1 | interferon regulatory factor 1 [Source:HGNC Symbol;Acc:6116] | protein coding | Pertussis Prolactin signaling pathway Hepatitis C Human papillomavirus infection |
| | | ENSG00000247275 | AL160008.1 | | lincRNA | |
| CCD229-002 | 2 | ENSG00000108984 | MAP2K6 | protein coding | protein coding | MAPK signaling pathway |
| | | ENSG00000152689 | RASGRP3 | RAS guanyl releasing protein 3 (calcium and DAGregulated) | protein coding | MAPK signaling pathway Ras signaling pathway Rap1 signaling pathway B cell receptor signaling pathway Pathways in cancer |

# Table 130: KEGG Pathways Enriched in Differentially Expressed Genes at Day 2 Compared to Pre-First Vaccination (RNA-Seq, Monocytes, Study Arm 1 A/H3N2v, D1)

Generate tables for each gene set category (KEGG Pathways, MSigDB Reactome Pathways, and MSigDB Immunologic Signatures), post-first vaccination day (Day 2, 4, 8, 29), Study Arm (Study Arm 1, 2, 3), all pairwise Study Arm Comparison (1 vs. 2, 1 vs. 3, 2 vs. 3), and cell type (monocytes, neutrophils, dendritic cells, NK cells B cell, and T cells). Repeat for post-second vaccination time points relative to pre-second vaccination for Study Arms 2 and 3.

| Gene Set ID | Gene Set<br>Genes # | Differentially Expressed Genes N (%) | Up-regulated Differentially<br>Expressed Genes N (%) | Down-regulated<br>Differentially Expressed<br>Genes N (%) | Jaccard Index | P-Value | FDR Adjusted P-<br>value |
|---|---|---|---|---|---|---|---|
| Influenza A | 62 | 9 (15) | 9 (15) | 0 | 0.234 | < 0.0001 | 0.0006 |
| Antigen processing and presentation | 59 | 4 (7) | 3 (5) | 1 (2) | 0.231 | <0.0001 | 0.0004 |

### 14.4 Safety Data

#### 14.4.1 Adverse Events

### 14.4.1.1 Adverse Events of Special Interest

Table 131: Number and Percentage of Subjects Experiencing Adverse Events of Special Interest

| | A/H3] | / Arm 1<br>N2v, D1<br>(=X) | A/H7N9 + A | Arm 2<br>AS03, D1, 29<br>=X) | Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) | |
|---|---|---|---|---|---|---|
| Category | n | % | n | % | n | % |
| Serious Adverse Event (SAE) | X | xx | x | XX | x | XX |
| Medically-Attended Adverse Event (MAAE) | X | xx | X | XX | X | xx |
| New-Onset Chronic Medical Condition (NOCMC) | X | xx | X | XX | X | xx |
| Potentially Immune-Mediated Medical Condition (PIMMC) | X | xx | X | XX | X | xx |
| N = Number of subjects in the Safety Analysis Population | | | | | | |

#### 14.4.1.2 **Solicited Adverse Events**

**Table 132:** Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, and Treatment **Group (Post-First Vaccination)** 

| | Study Arm 1<br>A/H3N2v, D1<br>(N=X) | | | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) | | | Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) | | |
|---|---|---|---|---|---|---|---|---|---|
| | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Any Symptom | x | XX | x x, x.x | X | XX | x x, x x | Х | XX | x x, x x |
| Any Systemic Symptom | х | XX | x x, x.x | Х | XX | x x, x x | Х | XX | x x, x x |
| [Systemic Symptom 1] | x | XX | x x, x.x | X | XX | x x, x x | Х | XX | x x, x x |
| [Systemic Symptom 2] | х | XX | x x, x.x | X | XX | x x, x x | Х | XX | x x, x x |
| Any Local Symptom | х | XX | x x, x.x | X | XX | x x, x x | X | XX | x x, x x |
| [Local Symptom 1] | х | XX | x x, x.x | X | XX | x x, x x | Х | XX | x x, x x |
| [Local Symptom 2] | х | XX | x x, x.x | X | xx | x x, x x | X | XX | x x, x x |

#### Tables with similar format:

Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, and Treatment **Table 133: Group (Post-Second Vaccination)** 

**Table 134:** Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, and Treatment **Group (Post-Any Vaccination)** 

Table 135: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group (Post-First Vaccination)

| | | | Study Arm 1<br>A/H3N2v, D1<br>(N=X) | | | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) | | | Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Any Symptom | None | Х | XX | x x, x.x | x | XX | x.x, x x | x | XX | x x, x.x |
| | Mild | Х | XX | x x, x.x | x | XX | x.x, x x | х | XX | x x, x.x |
| | Moderate | Х | XX | x x, x.x | х | XX | x.x, x x | х | XX | x x, x.x |
| | Severe | Х | XX | x x, x.x | х | XX | x.x, x x | х | XX | x x, x.x |
| Systemic Symptoms | | | | | | | | | | |
| Any Systemic Symptom | None | Х | XX | x x, x.x | х | XX | x.x, x x | х | XX | x x, x.x |
| | Mild | Х | XX | x x, x.x | x | XX | x.x, x x | X | XX | x x, x.x |
| | Moderate | X | XX | x x, x.x | X | XX | x.x, x x | X | XX | x x, x.x |
| | Severe | X | XX | x x, x.x | x | XX | x.x, x x | X | XX | x x, x.x |
| [Systemic Symptom 1] | None | X | XX | x x, x.x | X | XX | x.x, x x | X | XX | x x, x.x |
| | Mild | X | XX | x x, x.x | X | XX | x.x, x x | X | XX | x x, x.x |
| | Moderate | X | XX | x x, x.x | x | XX | x.x, x x | X | XX | x x, x.x |
| | Severe | Х | XX | x x, x.x | x | XX | x.x, x x | X | XX | x x, x.x |
| [Systemic Symptom 2] | None | Х | XX | x x, x.x | х | XX | x.x, x x | х | XX | x x, x.x |
| | Mild | Х | XX | x x, x.x | x | XX | x.x, x x | X | XX | x x, x.x |
| | Moderate | Х | XX | x x, x.x | x | XX | x.x, x x | X | XX | x x, x.x |
| | Severe | Х | XX | x x, x.x | X | XX | x.x, x x | X | XX | x x, x.x |
| Local Symptoms | | | | | _ | | | | | |
| Any Local Symptom | None | Х | XX | x x, x.x | х | XX | x.x, x x | х | XX | x x, x.x |
| | Mild | Х | XX | x x, x.x | х | XX | x.x, x x | х | XX | x x, x.x |
| | Moderate | Х | XX | x x, x.x | х | XX | x.x, x x | х | XX | x x, x.x |
| | Severe | X | XX | x x, x.x | X | XX | x.x, x x | X | XX | x x, x.x |

| | | | Study Arm 1<br>A/H3N2v, D1<br>(N=X) | | A/H | Study Arm 2<br>7N9 + AS03, I<br>(N=X) | | A/H | Study Arm 3<br>7N9 + PBS, D<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| [Local Symptom 1] | None | х | xx | x x, x.x | Х | xx | x.x, x x | X | xx | x x, x.x |
| | Mild | Х | xx | x x, x.x | х | xx | x.x, x x | X | xx | x x, x.x |
| | Moderate | Х | xx | x x, x.x | х | xx | x.x, x x | X | xx | x x, x.x |
| | Severe | Х | xx | x x, x.x | х | xx | x.x, x x | X | xx | x x, x.x |
| [Local Symptom 2] | None | Х | xx | x x, x.x | X | xx | x.x, x x | X | XX | x x, x.x |
| | Mild | Х | xx | x x, x.x | х | xx | x.x, x x | X | xx | x x, x.x |
| | Moderate | х | xx | x x, x.x | Х | xx | x.x, x x | х | xx | x x, x.x |
| | Severe | Х | xx | x x, x.x | Х | XX | x.x, x x | X | xx | x x, x.x |

 $N = Number\ of\ subjects\ in\ the\ Safety\ Analysis\ Population\ who\ received\ the\ specified\ dose.$ 

Severity is the maximum severity reported over all solicited symptoms post dosing for each subject.

#### Tables with similar format:

- Table 136: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group (Post-Second Vaccination)
- Table 137: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, and Treatment Group (Post-Any Vaccination)

Table 138: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Post-Vaccination Day (Post-First Vaccination, Study Arm 1 A/H3N2v, D1)

| | | | | | | | Study A | Arm 1 A/ | H3N2v, I | 01 (N=X) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | | re-<br>nation 1 | | ost-<br>nation 1 | Da | ay 1 | Da | ny 2 | Da | ny 3 | Da | ny 4 | Da | ny 5 | Da | у 6 | Day | y 7+ |
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any<br>Symptom | None | Х | XX | Х | XX | х | XX | х | XX | х | xx | х | XX | х | xx | х | xx | Х | XX |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Systemic Sym | nptoms | • | • | • | | | | | | | | | | | | | | | |
| Any<br>Systemic<br>Symptom | None | х | XX | Х | XX | х | XX | X | xx | Х | XX | Х | xx | Х | XX | Х | XX | X | xx |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| [Systemic<br>Symptom 1] | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| [Systemic<br>Symptom 2] | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |

| | | | | | | | Study A | Arm 1 A/1 | H3N2v, I | 1 (N=X) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | | re-<br>nation 1 | | ost-<br>nation 1 | Da | ny 1 | Da | y 2 | Da | ny 3 | Da | ny 4 | Da | ny 5 | Da | ny 6 | Day | y 7+ |
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Local Sympto | oms | | | | | | | | | | | | | | | | | | |
| Any Local<br>Symptom | None | х | xx | х | XX | х | XX | Х | xx | Х | xx | х | xx | х | XX | х | xx | х | XX |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| [Local<br>Symptom 1] | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| [Local<br>Symptom 2] | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |

N = Number of subjects in the Safety Analysis Population who received the specified dose. Severity is the maximum severity reported post dosing for each subject for each day.

#### Tables with similar format:

- Table 139: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Post-Vaccination Day (Post-First Vaccination, Study Arm 2 A/H7N9 + AS03, D1, 29)
- Table 140: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Post-Vaccination Day (Post-First Vaccination, Study Arm 3 A/H7N9 + PBS, D1, 29)
- Table 141: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Post-Vaccination Day (Post-Second Vaccination, Study Arm 2 A/H7N9 + AS03, D1, D29)
- Table 142: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, and Post-Vaccination Day (Post-Second Vaccination, Study Arm 3 A/H7N9 + PBS, D1, 29)

#### 14.4.1.3 Unsolicited Adverse Events

Table 143: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA® System Organ Class and Preferred Term, and Treatment Group (Post-First Vaccination)

| MedDRA® System Organ Class | MedDRA®<br>Preferred<br>Term | | Study Arm 1<br>A/H3N2v, D1<br>(N=X) | | A/E | Study Arm 2<br>17N9 + AS03, I<br>(N=X) | | A/I | Study Arm 3<br>H7N9 + PBS, D<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Any SOC | Any PT | Х | XX | xx, xx | Х | xx | xx, xx | х | XX | xx, xx |
| [SOC 1] | Any PT | | | | | | | | | |
| | [PT 1] | | | | | | | | | |
| | [PT 2] | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | |
| | [PT 1] | | | | | | | | | |
| | [PT 2] | | | | | | | | | |

Note: N = number of subjects in the Safety Analysis Population who received the specified dose. This table presents number and percentage of subjects. A subject is only counted once per PT.

#### Tables with similar format:

Table 144: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA® System Organ Class and Preferred Term, and Treatment Group (Post-Second Vaccination)

Table 145: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events with 95% Confidence Intervals by MedDRA® System Organ Class and Preferred Term, and Treatment Group (Post-Any Vaccination)

Table 146: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Maximum Severity, and Relationship (Study Arm 1 A/H3N2v, D1)

| | Study Arm 1 A/H3N2v, D1 (N=X) | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA® System Organ Class | MedDRA® Preferred Term | Any In | ıcidence | | | Sever | ity [1] | | | Re | elationship to | Treatment | [2] |
| | | | Mild Moderate Severe | | | | | ere | Not R | Related | Rel | ated | |
| | | n | % | n | % | n | % | n | % | n | % | n | % |
| Any SOC | Any PT | х | xx | Х | XX | х | XX | х | XX | х | xx | х | xx |
| [SOC 1] | Any PT | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | |

Note: N = Number of subjects in the Safety Analysis Population.

#### Tables with similar format:

Table 147: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Maximum Severity, Relationship (Study Arm 2 A/H7N9 + AS03, D1, 29)

Table 148: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Maximum Severity, Relationship (Study Arm 3 A/H7N9 + PBS, D1, 29)

<sup>[1]</sup> For severity, a subject is counted once per preferred term and is summarized according to their highest severity.

<sup>[2]</sup> For relationship, a subject is only counted once per preferred term and is summarized according to their closest relationship.

### 14.4.2 Listing of Deaths, Other Serious and Significant Adverse Events

### **Table 149:** Listing of Serious Adverse Events

| Adverse<br>Event | Associated with Dose # | # of Days Post Associated Dose (Duration) | # of Days<br>Post Dose<br>the Event<br>Became<br>Serious | Reason<br>Reported as<br>an SAE | Severity | Relationship<br>to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinue<br>d Due to<br>AE | Outcome | MedDRA®<br>System<br>Organ<br>Class | MedDRA®<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID: , | Treatment Gro | up: , AE Numb | er: | | | | | | | | | |
| Comments: | | | | | | | | | | | | |
| Subject ID: , | Treatment Gro | oup: , AE Numb | er: | | | | | | | | | |
| Comments: | | | | | | • | | | | | | |

### Table 150: Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events

| Adverse Event | Associated with Dose # | # of Days Post<br>Associated<br>Dose<br>(Duration) | Severity | Relationship<br>to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA®<br>System Organ<br>Class | MedDRA®<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID: , Tro | eatment Group:, | AE Number: | | | | | | | | |
| Comments: | | | | | | | | | | |
| Subject ID: , Tro | eatment Group:, | AE Number: | | | | | | | | |
| Comments: | | | | | | | | | | |

## Table 151: Listing of Adverse Events of Special Interest

| Adverse Event | Vaccination<br>Received at<br>Time of Event? | No. of Days<br>Post<br>Vaccination | Duration of<br>Event | Severity | MedDRA<br>System Organ<br>Class | NOCMC | PIMMC | Relationship | Outcome |
|---|---|---|---|---|---|---|---|---|---|
| | Subject ID: , Stud | ly Group: , AE Nun | nber: | I | l | l | I | I | |
| | Comments: | | | | | | | | |
| | Subject ID: , Stud | ly Group: , AE Nun | nber: | | | | | | |
| | Comments: | | | | | | | | |

### 14.4.3 Narratives of Deaths, Other Serious and Significant Adverse Events

(not included in SAP, but this is a placeholder for the CSR)

### 14.4.4 Displays of Vital Signs

Table 152: Vital Signs by Assessment, Maximum Severity, Study Day, and Treatment Group – Any Assessment

| | | A/H3 | y Arm 1<br>N2v, D1<br>K=X) | A/H7N9 + | y Arm 2<br>AS03, D1, 29<br>H=X) | A/H7N9 + | Arm 3<br>PBS, D1, 29<br>=X) |
|---|---|---|---|---|---|---|---|
| Study Visit Day | Severity | n | % | n | % | n | % |
| Day -7 (Screening) | None | X | xx | x | xx | x | xx |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| | Missing | | | | | | |
| Day 1 (Pre-Vaccination 1) | None | X | xx | Х | xx | х | XX |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| | Missing | | | | | | |
| Day 29 (Post-Vaccination 1) | None | n/a | n/a | х | xx | х | xx |
| | Mild | n/a | n/a | | | | |
| | Moderate | n/a | n/a | | | | |
| | Severe | n/a | n/a | | | | |
| | Missing | n/a | n/a | | | | |
| Maximum Post-Vaccination 1 | None | x | xx | х | xx | х | xx |
| | Mild | | | | | | |
| | Moderate | | | | | | |
| | Severe | | | | | | |
| | Missing | | | | | | |

| | | Study Arm 1<br>A/H3N2v, D1<br>(N=X) | Study Arm 2<br>A/H7N9 + AS03, D1, 29<br>(N=X) | Study Arm 3<br>A/H7N9 + PBS, D1, 29<br>(N=X) |
|---|---|---|---|---|
| 1 | Maximum Post-Vaccination 1 indicates the maximum severity experienced b | y each subject at any time point post baseline, include | ling unscheduled assessments. | |

N = Number of subjects in the Safety Analysis Population.

#### **Concomitant Medications**

Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group **Table 153:** 

| WHO Drug Code<br>Level 1, Anatomic Group | WHO Drug Code<br>Level 2, Therapeutic Subgroup | A/F | dy Arm 1<br>I3N2v, D1<br>(N=X) | A/H7N9 + | y Arm 2<br>AS03, D1, 29<br>N=X) | A/H7N9 + | y Arm 3<br>· PBS, D1, 29<br>N=X) |
|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % |
| Any Level 1 Codes | Any Level 2 Codes | X | XX | x | XX | Х | XX |
| [ATC Level 1 - 1] | Any [ATC 1 – 1] | | | | | | |
| | [ATC 2 - 1] | | | | | | |
| | [ATC 2 - 2] | | | | | | |
| | [ATC 2 - 3] | | | | | | |
| [ATC Level 1 – 2] | [ATC 2 - 1] | | | | | | |
| | [ATC 2 - 2] | | | | | | |
| | [ATC 2 - 3] | | | | | | |

N = Number of subjects in the Safety Analysis Population n = Number of subjects reporting taking at least one medication in the specific WHO Drug Class.

### **APPENDIX 2. FIGURE MOCK-UPS**

### LIST OF FIGURES

| Figure 1: | CONSORT Flow Diagram | 94 |
|---|---|---|
| Figure 2: | Hemagglutination Inhibition GMTs and 95% CIs by Study Arm and Post-Vaccination Day | 94 |
| Figure 3: | Barplot of Subject-Level Hemagglutination Inhibition Results at Day 29 Post-Last Vaccination | 95 |
| Figure 4: | Median Fold Change in Fractalkine Concentration and Associated 95% CI by Study Arm and Post-Vaccination Day | 96 |
| Figure 5: | Radar Plot of Median Fold Change by Study Arm and Post-Vaccination Day | 96 |
| Figure 6: | Multivariate starplots of reference alignment statistics | 97 |
| Figure 7: | Multivariate PCA, MDS, and hierarchical clustering plots | 98 |
| Figure 8: | Reverse empirical cumulative distribution function plots to summarize the percentage of genes that pass a certain average LCPM expression cut off | 99 |
| Figure 9: | MA and Volcano plots | 100 |
| Figure 10: | DE gene overlap between post-first vaccination days (Study Arm 1, Day 2-29 post-first vaccination) | 101 |
| Figure 11: | Heatmap, Co-Expressed Gene Cluster Dendrograms, and Cluster Time<br>Trend Visualizations | 102 |
| Figure 12: | Pathway Enrichment Visualizations | 103 |
| Figure 13: | Maximum Severity of Solicited Systemic Symptoms per Subject by Day (Post-First Vaccination) | 105 |
| Figure 14: | Incidence of Unsolicited Adverse Events by MedDRA® System Organ Class and Severity | 106 |

#### 10.1 Disposition of Subjects

#### Figure 1: CONSORT Flow Diagram

#### 14.2 Immunogenicity Data

Immunogenicity Response Figures by Measure, Treatment/Vaccination, and Time Point

Figure 2: Hemagglutination Inhibition GMTs and 95% CIs by Study Arm and Post-Vaccination Day



Repeat for neutralizing antibodies. Include all study arms. Label study arms as: Study Arm 1 A/H3N2v, D1; Study Arm 2 A/H7N9 + AS03, D1, 29; Study Arm 3 A/H7N9 + PBS, D1, 29.

Figure 3: Barplot of Subject-Level Hemagglutination Inhibition Results at Day 29 Post-Last Vaccination



Repeat for neutralizing antibodies. Include all study arms. Label study arms as: Study Arm 1 A/H3N2v, D1; Study Arm 2 A/H7N9 + ASO3, D1, 29; Study Arm 3 A/H7N9 + PBS, D1, 29.

Figure 4: Median Fold Change in Fractalkine Concentration and Associated 95% CI by Study Arm and Post-Vaccination Day



Plot individual fold change observations using treatment group-specific symbols. Include Study Arm 1 A/H3N2v. Label study arms as: Study Arm 1 A/H3N2v, D1; Study Arm 2 A/H7N9 + ASO3, D1, 29; Study Arm 3 A/H7N9 + PBS, D1, 29. Repeat for GM-CSF, IFN-γ, IL-1b, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12p70, IL-13, IL-17A, IL-21, IL-23, ITAC, MIP 1a, MIP1b, MIP3a, TNF-alpha, IP-10, IFNa, IFNb.

Figure 5: Radar Plot of Median Fold Change by Study Arm and Post-Vaccination Day



Include Study Arm 1 A/H3N2v. Label study arms as: Study Arm 1 A/H3N2v, D1; Study Arm 2 A/H7N9 + ASO3, D1, 29; Study Arm 3 A/H7N9 + PBS, D1, 29. Include Fractalkine GM-CSF, IFN-γ, IL-1b, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12p70, IL-13, IL-17A, IL-21, IL-23, ITAC, MIP 1a, MIP1b, MIP3a, TNF-alpha, IP-10, IFNa, IFNb.

#### 14.3 Transcriptomics Data

### Figure 6: Multivariate starplots of reference alignment statistics

Each sample is depicted by a star. Each ray represents one of the reference alignments statistics. Ray length is globally scaled so that the respective maximum alignment statistic across all samples is 1 and the minimum is 0. Stars will be color-coded by Study Arm.



Figure 7: Multivariate PCA, MDS, and hierarchical clustering plots

Standardized LCPM distributions will be used as input for PCA (A), MDS (B, C), and hierarchical clustering (D, E). For MDS and hierarchical clustering, results will be provided for Euclidean (B, D) as well as 1-Spearman correlation distance (C, E).



## Figure 8: Reverse empirical cumulative distribution function plots to summarize the percentage of genes that pass a certain average LCPM expression cut off

The x-axis represents the  $\log_2$  count per million cut off for identifying lowly expressed genes. The y-axis shows the percentage of all genes with a minimum gene expression level across all study samples that exceeds the respective cut off. The grey box indicates the target range of genes to be selected (between 10,000 and 14,000 genes). The black vertical lines represent the actual cut off that would be selected.



#### Figure 9: MA and Volcano plots

The y-axis on the MA plot (left panel) represents the log<sub>2</sub> fold change for the respective treatment effect. The x-axis shows the average log<sub>2</sub> expression level. The y-axis on the Volcano plot (right panel) represents the  $-log_{10}$  adjusted p-value and the x-axis the log<sub>2</sub> fold change for the respective treatment effect. Each black dot represents a gene. In red: DE genes. Blue dashed line: fold change cut off. MA and Volcano plots will be generated for each post-vaccination day, study arm, and study arm comparison.



Generate MA and Volcano plots for each post-first vaccination day (Day 2, 4, 8 or 29), Study Arm (Study Arm 1, 2, or 3), and pairwise Study Arm Comparison (1 vs. 2, 1 vs. 3, or 2 vs. 3). Repeat for post-second vaccination time points (Day 30, 32, and 36) relative to pre-second vaccination for Study Arms 2 and 3.

## Figure 10: DE gene overlap between post-first vaccination days (Study Arm 1, Day 2-29 post-first vaccination)

This plot summarizes the DE gene overlap between post-vaccination days for all DE (shown to the right), for up-regulated DE genes (shown in the middle), and down-regulated DE genes (shown to the right). For example, in the left panel, the bottom left horizontal barplot labeled 'SDEG Set Size' shows the total number of DE genes per post-vaccination time point. The black circles in the matrix represent what would be the different Venn diagram spaces (unique and overlapping DE genes). Connected black circles indicate a certain intersection of post-vaccination days. In the left panel, the first vertical bar/column shows those DE genes that are unique to Day 6. The second shows those DE genes that are shared only between Day 6 and 7. The third are those DE genes that are shared between Days 6, 7, and 8, and so forth.



Generate this plot for each study arm post-first vaccination. Repeat for post-second vaccination time points (Days 30, 32, and 36) relative to pre-second vaccination for Study Arms 2 and 3.
# Figure 11: Heatmap, Co-Expressed Gene Cluster Dendrograms, and Cluster Time Trend Visualizations

Left: Heatmap of log<sub>2</sub> fold changes of DE genes color-coded by up/down-regulation. Center: Gene cluster dendrogram with bootstrap probabilities and identified co-expressed gene clusters. Right: Time trends for mean log<sub>2</sub> fold changes and associated 95% bootstrap CI of co-expressed gene clusters.



Left: Generate heatmaps for each post-first vaccination day (Day 2, 4, 8 or 29), Study Arm (Study Arm 1, 2, and 3) and pairwise Study Arm Comparison (1 vs. 2, 1 vs. 3, 2 vs. 3). Repeat for post-second vaccination time points (Days 30, 32, and 36) relative to pre-second vaccination for Study Arms 2 and 3.

Center: Generate gene cluster dendrograms for each fold change set (Day 2-29 post-first vaccination and Day 2-8 post-second vaccination).

Right: Generate cluster time trends for each cluster and fold change set (Day 2-29 post-first vaccination and Day 2-8 post-second vaccination).

#### Figure 12: Pathway Enrichment Visualizations

**Left:** Pathway map of a significantly enriched pathway color-coded by up/down–regulation of genes.

Center: Heatmap summarizing pathway enrichment across study arms and post-vaccination days. Cells are color-coded by enrichment score:  $-1 \times \log_{10}(\text{enrichment p-value})$ . Numbers in each cell represent the number of DE genes. Two numbers will be printed in each cell: 1) the number of up-regulated DE genes and the 2) the number of down-regulated DE genes per pathway.

**Right:** Protein-protein interaction network centered around proteins encoded by DE genes. Nodes will be labeled by corresponding gene name. Edges will represent experimentally determined (reported in  $\geq 2$  publications) binary protein-protein interactions or protein complex membership. Color and size of individual nodes will indicate the mean log2 fold change between conditions. Further details are provided as part of the legend within the figure.



Left: Generate KEGG pathway maps for each enriched KEGG pathway for each post-first vaccination day (Day 2, 4, 8 or 29), Study Arm (Study Arm 1, 2, and 3) and pairwise Study Arm Comparison (Study Arm 1 vs.

2, 1 vs. 3, 2 vs. 3). Repeat for post-second vaccination time points (Days 30, 32, and 36) relative to presecond vaccination for Study Arms 2 and 3.

Center: Summarize for each gene set category (KEGG Pathways, MSigDB Reactome Pathways, MSigDB GO Biological Process, MSigDB Immunologic Signatures, and Blood Transcription Modules), for each post-first vaccination day (Day 2, 4, 8 or 29), Study Arm (Study Arm 1, 2, and 3) and pairwise Study Arm Comparison (1 vs. 2, 1 vs. 3, 2 vs. 3). Repeat for post-second vaccination time points (Days 30, 32, and 36) relative to presecond vaccination for Study Arms 2 and 3.

Right: Generate protein-interaction networks for H7N9 Study Arm Comparisons (Study Arm 1 vs. 2).

#### 14.4 Safety Data

Figure 13: Maximum Severity of Solicited Systemic Symptoms per Subject by Day (Post-First Vaccination)



Repeat for post-second vaccination and for solicited local symptoms. Include all study arms. Label study arms as: Study Arm 1 A/H3N2v, D1; Study Arm 2 A/H7N9 + ASO3, D1, 29; Study Arm 3 A/H7N9 + PBS, D1, 29.

Figure 14: Incidence of Unsolicited Adverse Events by MedDRA® System Organ Class and Severity



Include all study arms. Label study arms as: Study Arm 1 A/H3N2v, D1; Study Arm 2 A/H7N9 + ASO3, D1, 29; Study Arm 3 A/H7N9 + PBS, D1, 29.

# APPENDIX 3. LISTINGS MOCK-UPS

# **LISTINGS**

| Listing 1: | 16.1.6 Listing of Subjects Receiving Investigational Product | 109 |
|---|---|---|
| Listing 2: | 16.2.1 Early Terminations or Discontinued Subjects | |
| Listing 3: | 16.2.2.1 Subject-Specific Protocol Deviations | |
| Listing 4: | 16.2.2.2 Non-Subject-Specific Protocol Deviations | |
| Listing 5: | 16.2.3 Analysis Populations Exclusions | |
| Listing 6: | 16.2.4.1 Demographic Data | 114 |
| Listing 7: | 16.2.4.2 Pre-Existing and Concurrent Medical Conditions | 115 |
| Listing 8: | 16.2.6 Individual Immunogenicity Response Data – Antibody Assays | 116 |
| Listing 9: | 16.2.6 Individual Immunogenicity Response Data – Cytokine/Chemokine Assay | 116 |
| Listing 10: | 16.2.7.1 Solicited Events – Systemic Symptoms | |
| | 16.2.7.2 Solicited Events – Local Symptoms | |
| Listing 12: | 16.2.7.3 Unsolicited Adverse Events | 119 |
| Listing 13: | 16.2.9.1 Vital Signs | 120 |
| Listing 14: | 16.2.9.2 Physical Exam Findings | 120 |
| Listing 15: | 16.2.10 Concomitant Medications | 121 |

# Listing 1: 16.1.6 Listing of Subjects Receiving Investigational Product

| Subject ID | Randomized<br>Study Group | Product Received Study Vaccination 1 | Product Received Study Vaccination 2 |
|---|---|---|---|

#### 16.2 Database Listings by Subject

#### **16.2.1 Discontinued Subjects**

# **Listing 2:** 16.2.1 Early Terminations or Discontinued Subjects

| Treatment Group | Subject ID | Category | Reason for Early Termination or Treatment Discontinuation | Study Day |
|---|---|---|---|---|

#### **16.2.2 Protocol Deviations**

# **Listing 3:** 16.2.2.1 Subject-Specific Protocol Deviations

| Treatment<br>Group | Subject ID | DV Number | Deviation | Deviation<br>Category | Study Day | Reason for<br>Deviation | Deviation<br>Resulted<br>in AE? | Deviation Resulted<br>in Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|

# Listing 4: 16.2.2.2 Non-Subject-Specific Protocol Deviations

| Site | Start Date | Deviation | End Date | Reason for<br>Deviation | Deviation<br>Resulted in<br>Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Category | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|

# 16.2.3 Subjects Excluded from the Efficacy Analysis

#### Listing 5: 16.2.3 Analysis Populations Exclusions

| Treatment Group | Subject ID | Study Visit | Analyses in which<br>Subject is Included | Analyses from which<br>Subject is Excluded | Results Available? | Reason for Exclusion |
|---|---|---|---|---|---|---|
| | | | [e.g., Safety, ITT, PP] | [e.g., Safety, ITT, PP, Day x] | | |

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. "No" indicates that no data were available for inclusion in the analysis.

#### 16.2.4 Demographic Data

# Listing 6: 16.2.4.1 Demographic Data

| Treatment Group | Subject ID | Sex | Age at Enrollment (years) | Ethnicity | Race |
|---|---|---|---|---|---|

#### Listing 7: 16.2.4.2 Pre-Existing and Concurrent Medical Conditions

| Treatment<br>Group | Subject ID | MH Number | Medical History Term | Condition Start Day | Condition End Day | MedDRA System Organ Class | MedDRA Preferred Term |
|---|---|---|---|---|---|---|---|

#### 16.2.6 Individual Immunogenicity Response Data

Listing 8: 16.2.6 Individual Immunogenicity Response Data – Antibody Assays

| Treatment Group | Subject ID | Planned Time Point | Actual Study Day | HAI Titer | Neut Titer |
|---|---|---|---|---|---|

#### Listing 9: 16.2.6 Individual Immunogenicity Response Data – Cytokine/Chemokine Assay

| Treatment Group | Subject ID | Planned Time Point | Actual Study Day | Cytokine/Chemokine | Concentration |
|---|---|---|---|---|---|
| | | | | [Cytokine/Chemokine]* | |

<sup>\*:</sup> Fractalkine, GM-CSF, IFN-y, IL-1b, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12p70, IL-13, IL-17A, IL-21, IL-23, ITAC, MIP 1a, MIP1b, MIP3a, TNF-alpha, IP-10, IFNa, IFNb

#### 16.2.7 Adverse Events

#### **Listing 10:** 16.2.7.1 Solicited Events – Systemic Symptoms

| Treatment<br>Group | Subject ID | Dose Number | Post Dose Day | Assessmenta | Symptom | Severity | Attributed to<br>Alternate<br>Etiology? <sup>b</sup> | Alternate Etiology |
|---|---|---|---|---|---|---|---|---|
| | | | | MA | | | | |
| | | | | Clinic | | | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

<sup>&</sup>lt;sup>b</sup> Grade 3 events only.

**Listing 11:** 16.2.7.2 Solicited Events – Local Symptoms

| Treatment Group | Subject ID | Dose Number | Post Dose Day | Assessmenta | Symptom | Severity |
|---|---|---|---|---|---|---|
| | | | | MA | | |
| | | | | Clinic | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

#### Listing 12: 16.2.7.3 Unsolicited Adverse Events

| Adverse<br>Event | Associated with Dose No. | No. of Days Post Associated Dose (Duration) | Severity | SAE? | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment ( | Group: , Subject | ID: , AE Numbe | er: | • | • | | | | | | |
| Comments: | Comments: | | | | | | | | | | |
| Treatment ( | Group: , Subject | ID: , AE Numbe | er: | 1 | .1 | <u> </u> | <u> </u> | <u>l</u> | | <u> </u> | |
| Comments: | Comments: | | | | | | | | | | |
| Note: For a | dditional details | about SAEs, se | ee Table 149. | | | | | | | | |

#### 16.2.9 Vital Signs and Physical Exam Findings

#### Listing 13: 16.2.9.1 Vital Signs

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual Study<br>Day | Temperature<br>(°C) | Systolic Blood<br>Pressure<br>(mmHg) | Diastolic Blood<br>Pressure<br>(mmHg) | Heart Rate (beats/min) | Respiratory Rate (breaths/min) | Weight (kg) | Height (cm) |
|---|---|---|---|---|---|---|---|---|---|---|

# Listing 14: 16.2.9.2 Physical Exam Findings

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual Study<br>Day | Body System | Abnormal Finding | Reported as an AE?<br>(AE Description; Number) |
|---|---|---|---|---|---|---|

#### **16.2.10** Concomitant Medications

# **Listing 15:** 16.2.10 Concomitant Medications

| Treatment<br>Group | Subject ID | CM<br>Number | Medication | Medication Start<br>Day | Medication End<br>Day | Indication | Taken for an AE?<br>(AE Description;<br>Number) | Taken for a condition<br>on Medical History?<br>(MH Description;<br>Number) | ATC Level 1<br>(ATC Level 2) |
|---|---|---|---|---|---|---|---|---|---|